


# STATISTICAL ANALYSIS PLAN

# 2015-012-00US01

A Multi-Center, Open-Label, Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Surufatinib (HMPL-012), Previously Named Sulfatinib in Advanced Solid Tumors

AUTHOR: PPD

VERSION NUMBER AND DATE: V2.2, 04NOV2022




# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V2.2 (Dated 04NOV2022) for Protocol 2015-012-00US1 V7.0.

| | Name | Signature | Date |
|-----------|-------|-----------|------|
| Author: | PPD | PPD | |
| Position: | PPD | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|--------------|---------------------------|-----------|------|
| Approved By: | PPD | PPD | |
| Position: | PPD | | |
| Company: | IQVIA | | |
| Approved By: | PPD | PPD | |
| Position: | PPD | | |
| Company: | Hutchison Medi Pharma Ltd | | |


# MODIFICATION HISTORY

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| 0.1 | 25Feb2016 | PPD | Not Applicable – First Version |
| 0.2 | 17Mar2016 | PPD | Updated per sponsor's comments. Details can be found in the track change version. Additionally, following updates performed based on email communication: 1. ECG part added 2. Baseline definition added ECG time-point consideration 3. Subject disposition table modified to include completion status of DLT observation window. 4. Note added to explain EoT visit tumor assessment will contribute to all efficacy endpoints |
| 0.3 | 26Apr2016 | PPD | According to sponsor's comments, updated RECIST related details regarding tumor response confirmation are added to the SAP. One additional update regarding 2 or more missing consecutive visits' impact on PFS. Added Lab parameters grading according to CTC-AE guideline. |
| 0.4 | 30Sep2016 | PPD | Update comments. Update TLF according to new CRF. Add descriptions in SAP for each TLF. Previously, some TLFs don't have corresponding description in SAP. Revise layout |
| 0.5 | 24Nov2016 | PPD | Update comments |




| | | | "Shift Table of Laboratory Grade from Baseline" is replaced by "Shift in Toxicity Grading from Baseline to Worst CTCAE Grade" Add figures for QTcF and QTcB Merge lesion listings Merge some laboratory listings Remove or merge some tables to control the number of TLFs |
|---|---|---|---|
| 0.6 | 15Feb2017 | PPD | Update comments Update table "TEAEs by Severity" to have severity presented under each SOC/PT Combine table for "overall response" and "ORR and DCR" Remove table for DoOR and PFS Update derivation for exposure in Section 14.1 to more general description as new formulation, 200mg, is used. |
| 0.7 | 31JUL2017 | PPD | <ol> <li>Update while preparing dry run outputs</li> <li>Drop ATC 2nd level as ATC coding is not used for the study.</li> <li>Add baseline flags for data listings</li> <li>Move(add) definition for response evaluable set to section 6 for clear understanding</li> <li>Update section for ECG (external data)</li> <li>Update/modify table shells, especially ECG and laboratory parameters.</li> </ol> |
| 0.8 | 13May2019 | PPD | <ol> <li>Updated study title.</li> <li>Updated study primary objective and secondary objective.</li> <li>Updated study design.</li> <li>Updated definition of DLT evaluable patients.</li> <li>Updated analysis population and protocol deviation.</li> </ol> |




| 0.9 | 28MAY2019<br>28JUN2019 | PPD PPD | Updated the total sample size in the dose escalation phase and dose expansion phases. Updated the number of investigational centers. Updated efficacy objectives and endpoints. Updated comments from Hutchison Updated comments from Hutchison |
|---|---|---|---|
| 1.1 | 01JUN2020 | PPD | <ol> <li>Updated study title.</li> <li>Updated primary and secondary objectives and endpoints description based on protocol version 6.0 (Amendment 10).</li> <li>Updated the number of patients to be enrolled.</li> <li>Added sarcoma analysis description.</li> <li>Updated description for exploratory endpoints.</li> </ol> |
| 2.0 | 01ЛЛГ2020 | PPD | Updated comments from Hutchison. Updated Appendix 2 AESI list. |
| 2.1 | 24AUG2020 | PPD | Updated the definition of DLT evaluable patient per sponsor's note to file on 17Aug2020. Added the definition of treatment-emergent adverse event (TEAE). |
| 2.2 | 04NOV2022 | PPD | <ol> <li>Updated the Appendix 2 AESI list.</li> <li>Updated the protocol version as 7.0 (Amendment 11)</li> <li>Updated the MedDRA and WHO-DDE version</li> <li>Updated descriptions based on the wording changes in protocol version 7.0 (Amendment 11)</li> <li>Added additional analysis items for ECG in section 4.4</li> <li>Updated section 16.1.2 for BOR and add unconfirmed CR and PR for BOR</li> </ol> |





# TABLE OF CONTENTS

| 1. | LIST OF ABBREVIATIONS | 9 |
|------|------------------------------------------------------|----|
| 2. | INTRODUCTION | 12 |
| 3. | STUDY OBJECTIVES | 12 |
| 3.1. | | |
| 3. | 1.1. Primary Objective | |
| | 1.2. Secondary Objectives | |
| 3.2. | Dose Expansion Phase | |
| | 2.1. Primary Objective | |
| 3. | 2.2. Secondary Objectives | |
| 3. | 2.3. Exploratory Objective | |
| 4. | STUDY DESIGN | 14 |
| 4.1. | General Description | 14 |
| 4. | 1.1. Dose Escalation Phase | 14 |
| 4. | 1.2. Dose Expansion Phase | 15 |
| 4.2. | Sample Size | 10 |
| 4.3. | Schedule of Events | 17 |
| 4.4. | Changes to Analysis from Protocol | 17 |
| 5. | PLANNED ANALYSES | 17 |
| 5.1. | | |
| 5.2. | | |
| 5.3. | | |
| 5.4. | 1 2 | |
| 6. | ANALYSIS SETS AND PROTOCOL DEVIATIONS | 18 |
| 6.1. | | |
| 6.2. | Safety Analysis Set (SAS) – (All Treated Population) | |
| 6.3. | | |
| 6.4. | | |
| 6.5. | | |
| 7. | GENERAL CONSIDERATIONS | 20 |
| 7.1. | | |
| 7.2. | | |
| | End of Treatment | 21 |




| 7.3.1. End of Study | 21 |
|-------------------------------------------------------------|----|
| 7.4. Retests, Unscheduled Visits and Early Termination Data | 21 |
| 7.5. Visit Windows Conventions | |
| 7.6. Statistical Tests | |
| 7.7. Common Calculations | |
| 7.8. Software Version | 22 |
| 8. STATISTICAL CONSIDERATIONS | 27 |
| 8.1. Multicenter Studies | |
| 8.2. Missing data | |
| 9. OUTPUT PRESENTATIONS | 24 |
| 10. DISPOSITION AND WITHDRAWALS | |
| 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 11.1. Derivations | |
| 12. MEDICAL HISTORY AND ONCOLOGY HISTORY | |
| 12.1. Derivations | 29 |
| 13. MEDICATIONS AND PROCEDURES | 20 |
| 14. ONCOLOGY THERAPIES | |
| 15. STUDY MEDICATION EXPOSURE | |
| 15.1 DERIVATIONS | |
| 16. EFFICACY OUTCOMES | 32 |
| 16.1. Efficacy Variable(s) & Derivation(s) | |
| 16.1.1. Progression-Free Survival | |
| 16.1.2. Best Overall Response | |
| 16.1.3. Objective Response Rate | |
| 16.1.4. Disease Control Rate | |
| 16.1.5. Time to Response | |
| 16.1.6. Duration of Objective Response | |
| 16.1.7. Percentage Change in Tumor Size | |
| 16.2. Primary Analysis of Efficacy Variable(s) | |
| 16.3. Exploratory Efficacy 16.3.1. Tumor Markers | |
| 16.3.2. Overall Survival | |
| 16.4. Sensitivity Analysis of Efficacy Variable(s) | |
| 10.1. Scientify rhanges of Lineary variable(s) | |
| 17. SAFETY OUTCOMES | 39 |
| 17.1 Adverse Events | 30 |




| 17.1.1. All TEAEs | 40 |
|------------------------------------------------------------------------|----|
| 17.1.2. TEAEs Leading to Discontinuation of Study Medication | |
| 17.1.3. TEAEs Leading to Study Medication Adjustment | 41 |
| 17.1.4. Serious TEAEs | 41 |
| 17.1.5. TEAEs Of Special Interest (TEAESI) | 42 |
| 17.1.6. Dose Limiting Toxicity (DLT) | 42 |
| 17.1.7. Deaths | 42 |
| 17.2. Laboratory Evaluations | 42 |
| 17.2.1. Laboratory Specific Derivations | 43 |
| 17.2.2. Laboratory Reference Ranges and Markedly Abnormal Criteria | 43 |
| 17.2.3. CTCAE Grading for Laboratory Data | 44 |
| 17.2.4. Liver Function Abnormality | 44 |
| 17.3. ECG Evaluations | 45 |
| 17.3.1. ECG Specific Derivations | 45 |
| 17.3.2. ECG Markedly Abnormal Criteria | 45 |
| 17.3.3. Analysis of QTc Change from Baseline (ΔQTc) | |
| 17.3.4. Analysis of the Relationship Between QT/QTc and RR at Baseline | |
| 17.4. Vital Signs | |
| 17.4.1. Vital Signs Specific Derivations | |
| 17.4.2. Vital Signs Markedly Abnormal Criteria | |
| 17.5. Physical Examination | |
| 17.6. Other Safety Assessments | 48 |
| 17.6.1. ECOG Performance Status | |
| 17.6.2. Echocardiogram | 48 |
| 18. REFERENCES | 49 |
| APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | 50 |
| IQVIA Output Conventions | 50 |
| Dates & Times | 50 |
| Spelling Format | 50 |
| Presentation of Treatment Groups | 50 |
| Presentation of Disease Cohort | 51 |
| Presenting Order | 51 |
| APPENDIX 2. ADVERSE EVENTS OF SPECIAL INTEREST | |


# 1. LIST OF ABBREVIATIONS

| Terms and Abbreviations | Definition |
|-------------------------|------------------------------------------------|
| ACS | Abnormal, clinically significant |
| AE | Adverse event |
| ALT | Alanine aminotransaminase |
| ANCS | Abnormal, not clinically significant |
| aPTT | Activated partial thromboplastin time |
| AST | Aspartate amino transaminase |
| ATC | Anatomical Therapeutic Chemical |
| BOR | Best overall response |
| BTC | Biliary tract cancers |
| CA 19-9 | Carbohydrate antigen 19-9 |
| CCr | Creatinine clearance |
| CEA | Carcinoembryonic antigen |
| CgA | Chromogranin A |
| CI | Confidence interval |
| CR | Complete response |
| CRF | Case report form |
| CTC | Common toxicity criteria |
| CTCAE | Common terminology criteria for adverse events |
| DBL | Database Lock |
| DBP | Diastolic blood pressure |
| DCR | Disease control rate |
| DILI | Drug-induced liver injury |
| DLT | Dose-limiting toxicity |
| DoR | Duration of Response |
| EAS | Efficacy analysis set |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |




| Terms and Abbreviations | Definition |
|-------------------------|----------------------------------------------|
| ENR | All patients enrolled set |
| epNETs | Extrapancreatic neuroendocrine tumors |
| ICF | Informed consent form |
| INR | International nonproprietary ratio |
| LEVF | Left ventricular ejection fraction |
| LMS | Leiomyosarcoma |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MTD | Maximum tolerated dose |
| NCI | National Cancer Institute |
| NE | Not evaluable |
| NSE | Neuron-specific enolase |
| ORR | Overall response rate |
| OS | Overall survival |
| PD | Progression of disease |
| PFS | Progression-free survival |
| PK | pharmacokinetic |
| pNET | Pancreatic neuroendocrine tumors |
| PR | Partial response |
| RP2D | Recommended phase II dose |
| PT | Preferred term (MedDRA) |
| PVNS | Pigmented villonodular synovitis |
| QTc | QT interval corrected |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Safety analysis set |
| SBP | Systolic blood pressure |
| SCr | Serum creatinine |




| Terms and Abbreviations | Definition |
|---|---|
| SD | Stable disease |
| SMQ | Standardized MedDRA queries |
| SOC | System organ class (MedDRA) |
| SRC | Safety review committee |
| STS | Soft tissue sarcoma |
| Surufatinib | International non-proprietary name assigned to sulfatinib by the World<br>Health Organization |
| TSH | Thyroid stimulating hormone |
| TEAE | Treatment-emergent adverse event |
| TEAESI | Treatment-emergent adverse event of special interest |
| TTR | Time to response |
| UPS | Undifferentiated pleomorphic sarcoma |
| VEGF | Vascular endothelial growth factor |
| WHO | World Health Organization |


# 2. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for Protocol 2015-012-00US1. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 7.0 (amendment 11) dated 19Mar2021.

The pharmacokinetics analysis plan will not be included in this document.

## 3. STUDY OBJECTIVES

#### 3.1. Dose Escalation Phase

#### 3.1.1. Primary Objective

The primary objective is to evaluate the safety and tolerability of surufatinib in patients with advanced solid tumors of any type, and to determine the maximum tolerable dose (MTD) and/or recommended phase II dose (RP2D). Primary Endpoint: The incidence of Dose Limiting Toxicities (DLTs) in each cohort. DLT is defined in Section 6.3.

## 3.1.2. Secondary Objectives

The secondary objectives are:

- To evaluate the pharmacokinetic (PK) characteristics of multiple-dose surufatinib and to investigate the
  metabolite profile of surufatinib in the plasma of patients with solid tumors.
- To evaluate the anticancer activity of surufatinib in patients with advanced solid tumors of any type according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

#### Secondary Endpoints

- PK parameters: refer to pharmacokinetics analysis plan for details. PK parameters are listed below...
  - Maximum plasma concentration (C<sub>max</sub>)
  - Time to reach maximum concentration (T<sub>max</sub>)
  - Terminal half-life (t<sub>1/2</sub>)
  - Area under the concentration-time curve in a selected time interval (AUC<sub>0-t</sub>)
  - Area under the concentration-time curve in the time interval from 0 to infinity (AUC<sub>0...</sub>)
  - Apparent clearance (CL/F)
  - Apparent volume of distribution (V<sub>z</sub>/F)
  - Mean residence time (MRT)
  - Accumulation index based on AUC


 The objective response rate (ORR), disease control rate (DCR), duration of response (DoR), progressionfree survival (PFS), and percentage change in tumor size from baseline according to RECIST Version 1.1.

#### 3.2. DOSE EXPANSION PHASE

#### 3.2.1. Primary Objective

The primary objective is to evaluate the anticancer activity of surufatinib at the recommended Phase 2 dose (RP2D) from the dose escalation phase, in patients with advanced biliary tract cancer (BTC), patients with advanced Pancreatic Neuroendocrine Tumors (pNETs), patients with locally advanced, unresectable, metastatic Extrapancreatic Neuroendocrine Tumors (epNETs), and patients with soft tissue sarcoma (STS) treated at a dose of 300 mg QD (ie, the MTD/RP2D was declared in Protocol Amendment 7). The RP2D in this trial is the same as the RP2D used in clinical trials in China.

#### Primary Endpoints

- Patients with BTC (Arm A): progression-free survival (PFS) at 16 weeks (according to RECIST V.1.1.)
- Patients with pNET (Arm B): PFS at 11months (according to RECIST V.1.1.)
- Patients with epNET (Arm C): PFS at 11months (according to RECIST V.1.1.)
- Patients with STS (Arm D): PFS at 4 months (according to RECIST V.1.1.)

#### 3.2.2. Secondary Objectives

#### The secondary objectives are:

- To evaluate the PK profile of multiple dose surufatinib in patients with advanced BTC, patients with advanced pNET, patients with advanced epNET, and patients with advanced STS.
- To evaluate the safety of surufatinib in patients with advanced BTC, patients with advanced pNET, patients with advanced epNET, and patients with advanced STS.
- To evaluate the anticancer activity of surufatinib in patients with advanced BTC, patients with advanced pNET, patients with advanced epNET, and patients with advanced STS.

#### Secondary Endpoints:

- Pharmacokinetic parameters, which include but are not limited to, C<sub>max</sub>, T<sub>max</sub>, first-order rate constant K<sub>el</sub>, AUC, t<sub>1/2</sub>, CL/F, V<sub>z</sub>/F, accumulation ratio, and dose proportionality between AUC and dose and C<sub>max</sub> and dose.
- Safety, as assessed by:
  - The frequency and severity of adverse events
  - Physical examination findings
  - Vital signs


- Laboratory test results (ie, hematology, chemistry panel, and urinalysis)
- 12-lead electrocardiogram
- Echocardiogram
- ORR, DCR, time to response (TTR), DoR, and percentage change in tumor size from baseline defined according to RECIST V 1.1.

## 3.2.3. Exploratory Objective

The exploratory objectives are:

- To assess selected tumor markers based on type of malignancy.
- To evaluate the Overall Survival (OS) in patients with advanced BTC and advanced STS.

#### Exploratory Endpoint

- Tumor markers may include, but are not limited to, serum CEA and CA 19-9 (patients with BTC)
  serum chromogranin A (CgA) and neuron-specific enolase (NSE) for patients with pNET and epNET;
  and VEGF for the BTC, pNET and epNET disease cohorts. Assessment of tumor markers will be
  performed within 28 days prior to the start of treatment with study drug (C1D1) and at each tumor
  assessment visit.
- OS limited to patients enrolled to the BTC and STS cohorts only.

# 4. STUDY DESIGN

#### 4.1. GENERAL DESCRIPTION

This is an open-label, multi-center clinical trial of surufatinib taken orally once daily (QD), and it consists of 2 phases: a dose escalation phase in patients with advanced solid tumors of any type, and a dose expansion phase in patients with advanced BTC (Arm A), advanced pNETs (Arm B), advanced epNETs (Arm C), or STSs (Arm D) for whom standard therapy either does not exist or has proven to be ineffective or intolerable.

Approximately 95-150 patients will be enrolled in this 2-phase study: 35 patients in the dose escalation phase and approximately 115 patients in the dose expansion phase. The two phases will be conducted as described below.

#### 4.1.1. Dose Escalation Phase

In this phase, a 3+3 design will be used. Enrollment of 35-40 patients was planned. As of Protocol Amendment 7, a total of 35 evaluable patients have been enrolled in the dose escalation phase. The trial was to evaluate 5 surufatinib dose levels at 50,100, 200, 300 and 400 mg on a QD dosing schedule.


The study conduct was to follow a 3+3 design, with the dose limiting toxicity (DLT) assessment window being Cycle 1, from Day 1 to Day 28. Detailed description of a 3+3 design can be found in protocol section 5.1.1.

In addition to the five dose levels, in the occasion where 2 or more DLTs were observed in the 6 evaluable patients at a given dose level, the dose escalation was to be halted. If this dose level is greater than or equal to 50% higher than the previous dose level, an intermediate dose level was to be evaluated for toxicity in the same manner as a 3+3 dose level. If the dose level was less than 50% higher than the previous dose level, additional patients were to be enrolled at the previous dose level, if necessary, to form a dose cohort of minimum 6 evaluable patients. The MTD is the highest dose reached with no more than 1 DLT among 6 evaluable patients.

Any patient who was considered non-evaluable for DLT as defined in protocol section 5.1.1 'Dose escalation phase' was to be replaced by an additional patient at that same dose level.

Safety monitoring and evaluation for dose escalation will be carried out by a Safety Review Committee (SRC) upon completion of the DLT observation period of each dose level.

Patients who have completed the DLT observation window (Cycle 1, day 1-28) and were deemed to be benefiting from surufatinib treatment could have been permitted, at the investigator's discretion, to continue with surufatinib treatment until disease progression, death, intolerable toxicity, pregnancy, or loss of benefit from the study drug. Intra-patient dose escalation to a higher dose that had been cleared was allowed if the sponsor and investigator both agreed.

The MTD/RP2D of surufatinib has been declared at 300 mg QD (Protocol Amendment 7).

## 4.1.2. Dose Expansion Phase

The expansion phase will evaluate the antitumor activity of surufatinib, and evaluate the safety and tolerability of surufatinib at the RP2D determined at the end of the dose escalation phase.

Approximately 115 additional patients will be enrolled into the 4 open-label treatment arms during this phase: at least 30 patients with advanced BTC that have progressed on standard first-line chemotherapy will be assigned to Arm A, at least 15 patients with advanced pNET that have progressed on either everolimus, sunitinib, or both will be assigned to Arm B, and at least 15 patients with advanced epNETs that have progressed on everolimus will be




assigned to Arm C, and at least 55 patients with STS will be assigned to Arm D.

The safety of all enrolled patients will be closely monitored from the time of the initial dose of investigational treatment until 30 days after the last treatment dose. Any SAEs that occur after the ICF is signed, but before the first dose of study drug is taken, should also be reported. All AEs will be graded in accordance with the NCI CTCAE v. 4.03.

Patients will receive surufatinib continuously by 28-day treatment cycles until disease progression (according to RECIST Version 1.1), death, intolerable toxicity, or at investigator's discretion that the patient can no longer benefit from the study treatment. Tumor assessments will be conducted according to RECIST v. 1.1 criteria at screening, Cycle 2 Day 1 and every 8 (±1) weeks thereafter. Confirmation of CR and PR is required at no less than 4-week intervals between the date of initial response/progression and the confirmation assessment date.

#### 4.2. SAMPLE SIZE

The total number of patients enrolled will depend on the number of dose escalations and the need to further characterize individual cohorts in the expansion phase.

Approximately 95-150 patients will be enrolled in this two-phase study: 35 patients in the dose escalation phase and approximately 115 additional patients in the dose expansion phase. The actual enrollment number may vary, depending on the number of dose levels evaluated and the number of DLTs observed in each cohort, as well as the potential need to further characterize individual cohorts in the dose expansion phase.

As per Protocol Amendment 7, an additional 15 patients will be enrolled into Arm A (BTC) of the expansion phase, for a total enrollment of at least 30 advanced BTC patients. The reason for increasing enrollment into Arm A (advanced BTC) is that preliminary data from the ongoing patients in this cohort have shown encouraging results. The additional patients will allow further characterization of the safety and efficacy of surufatinib in this patient population. Arm B (pNET) and Arm C (epNET) will enroll at least 15 patients each. If needed, Arm B and Arm C could enroll additional patients in order to characterize further the safety and efficacy of surufatinib in these patient populations.

As per Protocol Amendment 8, 45 patients with STS (10 patients with Leiomyosarcoma (LMS), 10 patients with Undifferentiated pleomorphic sarcoma (UPS), 10 patients with epithelioid sarcoma, 10 patients with angiosarcoma, 10 patients with synovial sarcoma, and 5 patients with Pigmented villonodular synovitis (PVNS)) are planned to be


enrolled.

As per Protocol Amendment 10, an additional 10 patients will be added to the arm D (STS) for a total enrolment of 55 patients.

Additional details on sample size can be found in Protocol Section 10.1.

#### 4.3. SCHEDULE OF EVENTS

Schedule of events can be found in Protocol Appendix 1 - Study Flowcharts.

#### 4.4. CHANGES TO ANALYSIS FROM PROTOCOL

Additional Analysis for ECG will be included the evaluation of change from baseline in QTcF ( $\Delta$ QTcF) intervals and the relationship between QT/QTc and RR intervals at baseline will be evaluated graphically. Refer to the section 17.3.3 and 17.3.4 for the details.

# 5. PLANNED ANALYSES

The following formal analyses are planned for the study:

## 5.1. SAFETY REVIEW COMMITTEE (SRC)

Safety monitoring and evaluation for dose escalation will be carried out by a Safety Review Committee (SRC) upon completion of the DLT observation period of each cohort.

The SRC is chaired by the Sponsor's Clinical Program Leader of the surufatinib program, and members will include the principal investigators (PIs), the Sponsor's PK scientist, medical monitor, and safety scientist, and the CRO's medical monitor. Dose escalation decisions are based on safety and PK data from this ongoing trial, as well as consideration of safety and PK data at comparable drug exposures from patients in previously conducted clinical trials in China.

For the dose expansion phase of the trial, a separate, specific SRC will be established to ensure the safety of all patients treated with study drug in the STS cohort (STS-SCR). Review of available safety laboratories, adverse events, and any other pertinent data available will be reviewed after the first 4 patients in each sarcoma cohort have completed at least 1 cycle of treatment. The recommendations of the STS-SRC will be based on the members'


clinical assessment of the cumulative safety data provided for review. The SRC will not be charged with the application of formal statistical stopping rules for safety.

#### 5.2. Interim Analysis

An informal interim analysis was performed using data cut-off date of 30JUN2020. This SAP covers the analyses for efficacy and safety based on the data cut-off for the interim analysis. The interim analysis was performed using cleaned eCRF data collected until data cut-off date. In addition, SAEs were be summarized based on all patients recruited into study on or before data cut-off date. All SAE data to be included in the interim analysis was to be cleaned.

Considering the goal of this interim analysis was to support regulatory submission, the efficacy analysis for this interim analysis was limited to pNET and epNET cohorts while the safety was cover all patients enrolled on the trial as of the planned cut-off date.

In addition, the overall survival analysis for BTC and STS cohorts were not included in this interim analysis. The tumor assessment after the end of treatment was not applied to this interim analysis as well. The tumor assessment data after the end of treatment was cut-off for this interim analysis.

#### 5.3. SNAP SHOT ANALYSIS

A snap shot analysis was performed using data at cut-off date of 14Jun2019.

All summaries of safety and efficacy data were presented by assigned dose level in escalation phase, and disease type which pooled the patients who enrolled in the dose expansion phase and patients of the same tumor type (BTC, pNET, epNET) at the RP2D dose level in the dose escalation phase.

# 5.4. FINAL ANALYSIS

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics by following sponsor's authorization of this SAP and final Database Lock (DBL) for this study.

# 6. ANALYSIS SETS AND PROTOCOL DEVIATIONS

Agreement and authorization of patients included/ excluded from each analysis set will be conducted prior to the


DBL for the final analysis of the study.

All summaries will be presented by assigned dose level in escalation phase, and by disease type which will pool the patients who enrolled in the dose expansion phase and patients of the same tumor type (BTC, pNET, epNET, STS) at the RP2D dose level in the dose escalation phase.

All patients will be presented according to their initial assigned dose level regardless of any dose adjustment during study conduct.

# 6.1. ALL PATIENTS ENROLLED SET [ENR]

The all patients enrolled set (ENR) will include all patients who signed informed consent form (ICF) for this study.

## 6.2. SAFETY ANALYSIS SET (SAS) – (ALL TREATED POPULATION)

This analysis set includes all patients who have received at least one dose of surufatinib. Safety data will be evaluated based on this analysis set outcome. Patients in the SAS will be analyzed by their actual dose initially received. If patients have dose reduction during the study, all data will be summarized/ analyzed based on the initial dose of study medication received.

All safety analyses except for DLT summaries will be based on the SAS. Efficacy endpoints PFS and OS (OS applies to BTC and STS cohorts only) will be analyzed based on this analysis set.

## 6.3. DOSING LIMITING TOXICITY (DLT) EVALUABLE SET

The DLT set comprises all SAS patients who are evaluable for DLT assessment. DLT evaluable patients can be identified via answers to the question "DLT evaluable patients" on CRF "DLT Assessment" page.

DLT set (and summaries of DLTs) only applies to dose escalation phase patients.

A DLT evaluable patient has to meet the following criteria, which will not be confirmed via programming:

- Has not received any preventive treatment during the DLT period; AND
- Has completed the first 28-day treatment cycle with complete safety evaluations and has received at least 75% of the assigned surufatinib dose; OR
- Has a confirmed DLT during the first 28-day treatment cycle.

#### 6.4. EFFICACY ANALYSIS SET (EAS)

This analysis set includes all patients who have received at least one dose of surufatinib and have had at least one


post-baseline tumor assessment.

All efficacy endpoints will be analyzed based on this analysis set except for analysis of PFS and OS, which will be analyzed based on the SAS. The OS analysis will be performed for the BTC and STS cohorts only.

#### 6.5. PROTOCOL DEVIATION

Major protocol deviations related to study inclusion or exclusion criteria, conduct of the trial, patient management, or patient assessment will be listed for SAS.

The study team will discuss, identify and classify the important eligibility criteria or post-entry deviations from operational team monitor reports before final data base lock.

# 7. GENERAL CONSIDERATIONS

## 7.1. REFERENCE START DATE, REFERENCE END DATE AND STUDY DAY

Reference start date is defined as the date of the first administration of study medication. Study day will be calculated from the reference start date and will be used to show start/stop day of the assessments and events relative to the first administration of study medication.

Reference end date will be defined as the day of the last administration of study medication within the patient's last treatment cycle.

Study day (Day 1 is the day of the first administration of study medication) will appear in each listing where an assessment date or event date appears.

If the date of the event is on or after the reference start date then:

Study day = (date of event - reference start date) + 1.

If the date of the event is prior to the reference start date then:

Study day = (date of event - reference start date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, Study day, and any corresponding durations will be presented based on the imputations specified in Section 8.2. In addition to the overall reference start and end date, the start and end of treatment within each cycle will be identified based on the data collected on the eCRF form and will be used when assigning events or assessments to a particular treatment cycle.




#### 7.2. BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In case where the last non-missing measurement and the reference start date coincide, that measurement will be considered as baseline, but AEs and medications commencing on the reference start date will be considered post-baseline, that is, treatment-emergent or concomitant ("worst case" approach).

#### 7.3. END OF TREATMENT

End of treatment reasons and treatment discontinuation date are captured on CRF page "End of Treatment". Patients who complete or prematurely discontinue the study medication need to return to the study site for a follow-up within 30±7 days after the last dose of surufatinib. Measurements obtained during this visit will be considered as the 'End of Treatment' assessment.

#### 7.3.1. End of Study

A patient is considered to have completed the study once he or she has completed the last visit, or the last scheduled procedure as outlined in the Schedule of Events in Protocol Appendix 1.

#### 7.4. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the nominal visit will be presented. Unscheduled measurements will not be included in by-visit summaries. Unscheduled measurements will contribute to worst-case summaries. In the case of a retest (visit-specific unscheduled visit number assigned), the latest non-missing measurement among all scheduled and unscheduled measurements for that visit will be used for by-visit summaries.

Early termination data of patients prematurely discontinued from study medication will be presented together with the end of treatment assessment for study medication completers.

By-parient listings will include scheduled, unscheduled, retest, and early discontinuation data.

#### 7.5. VISIT WINDOWS CONVENTIONS

Unless otherwise indicated, in the treatment period, during Cycle 1 and Cycle 2, the visit window will be  $\pm 1$  day. From Cycle 3 onward, the visit window will be  $\pm 3$  days. In the follow-up visit, the visit window is  $\pm 7$  days. All data will be organized and analyzed according to the scheduled times as outlined in the protocol and by the visit


denoted on the Case Report Form (CRF).

#### 7.6. STATISTICAL TESTS

There is no formal statistical hypothesis testing in this study. The confidence intervals will be 95%, unless otherwise specified in the description of the analyses.

#### 7.7. COMMON CALCULATIONS

For quantitative measurements, change from Baseline will be calculated as:

- Change from baseline = Test Value at Visit X Baseline Value
- Percentage change from baseline = [(Test Value at Visit X Baseline Value) / Baseline Value] \* 100

The time from Date of Event A to Date of Event B (years) is calculated as:

(Date of Event B - Date of Event A + 1)/365.25.

The time from Date of Event A to Date of Event B (months) is calculated as:

(Date of Event B - Date of Event A + 1)/30.4375.

#### 7.8. SOFTWARE VERSION

All analyses will be conducted using SAS® Version 9.4 or higher.

# 8. STATISTICAL CONSIDERATIONS

#### 8.1. MULTICENTER STUDIES

This study will be conducted by multiple investigators at approximately 8-15 sites. No adjustment in aspect of site effect will be performed. Data from all centers will be pooled prior to analysis.

#### 8.2. MISSING DATA

Generally, the missing efficacy and safety data will not be imputed except for the critical missing and incomplete dates which will be handled as described in this section.




For partially missing dates, the Age (Years), Duration of malignancy (years) and Duration of metastasis (years) will be based on imputed values. For all calculation elements, if the date part is missing while year and month present, 15<sup>th</sup> of the month will be used for imputation. If both date and month part are missing while year presents, July 1<sup>st</sup> will be used for imputation.

When no imaging/measurement was done at all at a particular time point, the patient is not evaluable at that timepoint. If only a subset of lesion measurements were made at an assessment, usually the case is also considered not evaluable at that timepoint, unless a convincing argument can be made that the contribution of the individual missing lesion(s) would not change the assigned time point response.

For ORR and DCR calculation, patients with missing responses will be considered non-responders, thus contribute only to the denominator.

#### Initial Diagnosis Date

If year and month are known but the day is unknown, day will be imputed as 15. If only year is known, month and day will be imputed to July 1st. If the diagnosis date is completely missing or the year part is unknown, the diagnosis date will not be imputed. The imputed date will be compared to reference start date. If it is later than the reference start date, the incomplete date will be imputed as the reference start date.

#### Adverse Events Date

For adverse event, incomplete start dates and/or stop dates will be imputed. Start date will be imputed first when the start date and stop date are both incomplete for a patient. If the field of year is missing, then no value will be imputed. The following rules will be applied to impute the incomplete start date, assuming year is available.

#### Missing or incomplete start date

In case the start date of an AE is completely missing, or year part is unknown, the start date of AE will not be imputed.

In case the start date of AE is in the same year as reference start date (when only year is recorded), or the start date is in the same month and year (if only the day is missing) as the reference start date, then the start date of the AE will be imputed by the minimum of the reference start date and the AE resolution date. In all other cases the available year and month are not equal to the corresponding year and month of the reference start date or the available year is not equal to the corresponding year of the reference start date, the missing start day will be imputed by the 1st day of the month and the missing start month will be replaced by January.

In the case only the month is missing while year and day are recorded, then both day and month will be considered as missing. If the year part of start date of an AE occurs in the same year as reference start date, then the start date of




the AE will be imputed by the minimum of the reference start date and the AE resolution date. If an AE is observed on different year of the reference start date, January 1st will be used to complete the start date of the AE..

#### Missing or incomplete end date

Incomplete end dates will be imputed to the last possible date. In the case the year and month are known, AE end date will be imputed as the last day of the month. In the case if only the year is known, AE end date will be imputed as the December 31<sup>st</sup> of the year. If the imputed AE end date is after the death date, then the date of the death will be imputed as the AE end date. If the end date is completely missing or the year part is unknown, the end date will not be imputed. If the imputed end date is before the start date (imputed or non-imputed start date), then the stop date will be imputed using start date.

For AE events continuing at the cut-off date, the end date will not be imputed and will be reported as "ongoing".

#### Medications/Procedures Date

There will be no imputation for complete missing start date or end date of medications/procedures.

Impute incomplete start date as earliest possible date, i.e. first day of month if day unknown or 1st January if day and month are unknown.

Impute end date as latest possible date, i.e. last day of month if day unknown or 31st December if day and month are unknown, if not resulting in a date later than the date of patient's death. In the latter case the date of the death will be used to impute the incomplete stop date.

Above rules will be applied for prior/concomitant medications/ procedures and prior oncology therapies.

Duration will not be calculated in case either the start date or end date is completely missing, but it will be calculated based on the imputed start/ end date if either the start date or end date is incomplete.

Last Tumor Assessment Date

If year and month are known but the day is unknown, day will be imputed as the first day of the month. If only year is known or a date is complete missing, the date will not be imputed. If the date of death is complete, the imputed date will be compared with the death date, the earlier date will be used for the date of last tumor assessment.

Subsequent Anti-tumor Therapy Date

When an incomplete subsequent anti-tumor therapy start date is reported, every effort will be made to identify the precedence relationship of starting date of subsequent anti-tumor therapy relative to the reference end date and the date of disease progression (if happened). Generally, records of subsequent therapy should all start after EOT/PD.


| | Condition | Reference end date<br>(D1) | Date of earliest disease<br>progression (D2) | Imputed start date for anti-<br>tumor therapy |
|---|---|---|---|---|
| Known part | 1 | Before | Before | Minimum (D1, D2) -1 |
| or clinical | 2 | After | After | Maximum (D1, D2) +1 |
| evidence to | 3 | Before | After | D2+1 |
| show | 4 | After | Before | D2-1 |
| precedence | 5 | No or not applicable | Before | D2-1 |
| relationship | 6 | No or not applicable | After or others | D2+1 |
| | 7 | Before | No or not applicable | D1-1 |
| | 8 | After or others | No or not applicable | D1+1 |

For example, condition 3, if the known part of the anti-tumor therapy indication that the anti-tumor therapy starts before reference end date but after date of disease progression, then incomplete start date of anti-tumor therapy will be imputed as one day posterior to date of disease progression.

If the imputed start date is later than date of death, then the imputed start date will be further imputed to date of death

#### Death Date

If year and month of death date are known but the day is unknown, day will be imputed as 15. If only year is known, month and day will be imputed to July 1st. There are two exceptions of the below two scenarios:

- If the imputed death date is prior to the last known alive date, then the death date will be imputed to the next day of last known alive date.
- If the imputed death date is after end of study date with the year and month are the same as end of study date, then the death date will be imputed to the date of end of study.

# 9. OUTPUT PRESENTATIONS

Appendix 1 details the conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures and listings to be provided by IQVIA Biostatistics.

Continuous variables will be summarized using descriptive statistics, i.e., number of patients(n), mean, median, standard deviation (SD), and ranges (minimum, maximum).

Qualitative variables will be summarized by count(s) and percentages (%). Unless otherwise stated, the calculation of percentages will be based on the total number of included in the relevant analysis set.


# 10. DISPOSITION AND WITHDRAWALS

All patients who signed ICF will be involved in the analysis of disposition and withdrawals being described in this section for this study.

The number of patients who signed ICF for the study, screen failed patients along with the reason for screen failure, patients who passed screening but withdraw before the first dose of study treatment will also be summarized. The number of patients included/excluded from each analysis set as well as the reason(s) for exclusion (as described in Section 6) will also be summarized by dose level in escalation phase and by disease cohort in dose expansion phase. A corresponding by-patient listing will also be provided.

The number and percentage of patients who completed, discontinued from study medication and reasons for study medication discontinuation will be presented for each dose level, by disease cohort, and overall for the SAS. Reasons for discontinuation of study medication will be presented as recorded on the CRF page "End of Treatment". The number and percentage of patients who completed, discontinued from study and reasons for study discontinuation will be presented for each dose level, disease cohort, and overall for the SAS. Reasons for study discontinuation will be presented as recorded on the CRF page "End of Study".

A patient listing will be generated to include site, patient number, informed consent information (date), screening date, first and last study medication dosing date, duration of study medication, study medication discontinuation information (date and reason), and end of study information (date, status, and reason for discontinuation if applicable) will be provided. Besides, the violation of inclusion/exclusion criteria will also be listed for ENR analysis set.

Major protocol deviations related to study inclusion or exclusion criteria, conduct of the trial, patient management, or patient assessment will be listed..

# 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be summarized by dose cohort in dose escalation phase and by disease cohort in dose expansion phase for the SAS. Data listing will also be provided.

The following demographic and other baseline characteristics will be reported and listed for this study:

- Age (years) Calculated relative to date of ICF
- Age group
  - <65 years</li>
  - ≥65 years
- Gender




- Male
- Female
  - With Child Bearing Potential
  - Without Child Bearing Potential
  - Undifferentiated
- Unknown

#### Race

- American Indian or Alaska Native
- Asian
- o Black or African American
- Native Hawaiian or Other Pacific Islanders
- White
- Other

#### Ethnicity

- Hispanic or Latino
- o Not Hispanic or Latino
- Not Reported
- Unknown
- Baseline Weight (kg)
- Baseline Height (m)
- Baseline BMI (kg/m²)
- Baseline ECOG performance status (refer Section 17.6.1)
  - 0 0
  - 0 1
  - o >1
- Baseline Sum of Diameters of Target Lesions (mm)

Other baseline characteristics related to the oncology history will be described in Section 12.


#### 11.1. DERIVATIONS

- BMI (kg/ m<sup>2</sup>) = weight (kg)/ height (m)<sup>2</sup>
- Age (Years) = (Date of Informed Consent Signed Date of Birth + 1)/365.25

# 12. MEDICAL HISTORY AND ONCOLOGY HISTORY

Pre-existing medical conditions are recorded on the "Medical History" CRF page.

Medical history (excluding oncology history) will be summarized by system organ class (SOC) and preferred term (PT) for the SAS set. Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary, Version 23.0 (MedDRA 23.0) or higher will be used for coding. Number and percentage will be presented in frequency tables by dose cohort in dose escalation phase and disease cohort in dose expansion phase, and ordered by primary SOC and PT in descending order of the frequency in total within each category. For SOCs or PTs with the same frequency in total, categories will be sorted alphabetically.

Oncology history information will be captured on CRF page "Oncology History" and the following oncology history information will be summarized:

- Type of malignancy
- Duration of malignancy (years) Calculated relative to date of ICF
- Time since the initial diagnosis to first administration of study medication (years) Calculated relative to date of first administration of study medication
- Stage of the disease at the time of initial diagnosis
  - Stage I
  - Stage II
  - Stage III
  - Stage IV
- Metastasis Status (Yes, No)
- Duration of Metastasis (Years) Calculated relative to date of ICF
- Prior oncology treatments
  - Oncology Chemotherapy and Medication
  - Oncology Radiation Therapy
  - Oncology Surgery and Procedures

Medical history and oncology history will be listed for the SAS.


#### 12.1. DERIVATIONS

- Duration of malignancy (years) = (Date of Informed Consent Signed Date of first confirmed malignancy + 1)/365.25.
- Time since the initial diagnosis to first administration of study medication (years) = (Date of first administration of study medication – Initial primary diagnosis date for solid tumor + 1)/365.25.
- Duration of metastasis (years) = (Date of Informed Consent Signed Date of metastasis observed + 1)/365.25.

# 13. MEDICATIONS AND PROCEDURES

Prior medications are medications which ended prior to the first dosing date of study medication. Concomitant medications/procedures are medications/procedures which started no later than 30+7 days following the last dose administration, and ended on or after the date of first dose of medication or were ongoing at the end of the study. Relevant information is collected on CRF page "Prior and Concomitant Medications", "Concomitant Procedures". Prior and concomitant medications will be coded using World Health Organization Drug Dictionary Enhanced (WHO-DDE), version Mar2020 or latest version. Anatomical Therapeutic Chemical (ATC) level 2 classification and Preferred term (PT) will be used for coding.

Concomitant medications will be summarized by ATC level 2 and PT for each dose cohort in dose escalation phase and each disease cohort in dose expansion phase for the SAS. PT will be sorted in descending frequency of the total number of patients with at least one medication in the corresponding category, PTs will be presented alphabetically for PTs of the same total frequency.

Concomitant procedures will be coded by MedDRA 23.0 or higher and will be presented by PT by dose cohort in dose escalation phase and by disease cohort in dose expansion phase. PT will be sorted in descending frequency of the total number of patients with at least one procedure in the corresponding category, PTs will be presented alphabetically for PTs of the same total frequency.

Prior and concomitant medications will be presented in listings with flag to differentiate whether the medication was prior medication or concomitant medication. Similar for prior and concomitant procedures information.

# 14. ONCOLOGY THERAPIES

Prior oncology therapies include oncology chemotherapy and medication, oncology radiotherapy, and oncology surgery and procedures. Oncology chemo therapy and medication will be captured on "Oncology Chemotherapy and




Oncology Medication" CRF page, oncology radiotherapy will be captured on "Oncology Radiotherapy" CRF page, and oncology surgery and procedures will be captured on "Oncology Surgery and Procedure" CRF page. Prior oncology chemotherapies and medications will be coded using WHO-DDE, version Mar2020 or latest version, and will be presented by ATC level 2 classification and PTs for each dose cohort in dose escalation phase and each disease cohort in dose expansion phase for the SAS. PT will be sorted in descending frequency of the total number of patients with at least one condition in the corresponding category, PTs will be presented alphabetically for PTs of the same total frequency. In addition, number and percentage of patients who received prior oncology chemotherapies and medications, number of regimens, best response, treatment failure information and appearance of adverse reaction with severity above grade 3 will be summarized for prior oncology chemotherapies and medications.

The number and percentage of patients who received prior oncology radiotherapy, purpose, best response, and appearance of adverse reaction with severity above grade 3 will be summarized for prior oncology radiotherapy. Prior oncology surgery and procedure will be coded using MedDRA 23.0 or higher, and will be summarized by SOC and PT for each disease cohort in dose expansion phase and dose escalation phase for the SAS. SOC and PT will be sorted in descending frequency of the total number of patients with at least one condition in the corresponding category, SOCs/PTs will be presented alphabetically for SOCs/PTs of the same total frequency. Since on-study oncology therapies are not allowed, oncology therapies will be classified and reported as prior. Any concurrent oncology therapy will be considered and reported as protocol deviation.

. All the oncology therapies as well as general therapies will be listed by disease cohort in dose expansion phase and dose escalation phase.

Oncology chemotherapy and oncology medication, oncology radiotherapy, and oncology surgery and procedure will be listed for SAS. Oncology surgery and procedure will be listed for SAS and will be presented separately from concomitant procedures.

New anti-tumor therapy is defined as any anti-tumor therapy started after first dose of study medication. New antitumor therapy will be flagged in the listing of oncology medication/radiotherapy/surgery.

# 15. STUDY MEDICATION EXPOSURE

The extent of exposure to study medication will be presented by dose cohort and disease cohort for cycle 1 (DLT window) and overall respectively for the SAS.

Study medication exposure calculation will be based on study medication administration information, which is collected on the CRF pages "Study Drug Administration". In the case of missing data on the eCRF or if derivations are required, the "Study Drug Administration" or "Study Drug Dispensation and Return" form will be used in order


to determine the first and the last date of study medication.

Descriptive information will be provided regarding number of cycles exposure to study drug, total duration of study medication exposure, actual duration of study medication taken, cumulative dose of study medication, dose intensity and relative dose intensity as both continuous variable and categorical variable (<80%, >=80% and <=120%,

>120%). The number and percentage of patients with any prescribe dose increased, reductions and interruptions will be presented, the timing of prescribe dose increased, reductions and interruptions and reasons for dose increased, reductions and interruptions will be summarized as well.

Additionally, the relative dose intensity calculated for DLT observation window (28 days since first dose regardless of the actual date of C2D1 visit) will facilitate the determination of DLT set and will be presented together in a listing with overall study medication exposure.

Study medication administration in each cycle will be taken from CRF page "Study Drug Administration" at each visit.

Study drug administration data will be listed by dose cohort in dose escalation phase and by disease cohort in dose expansion phase. And any dose modifications will be flagged.

Another listing of study medication accountability with relevant information will be provided.

# 15.1 DERIVATIONS

- Total duration of study medication (Days) in cycle 1= Stop date of administration in cycle 1 Start date of administration +1
- Total duration of study medication (Days) for overall = Stop date of administration in last cycle Start date
  of administration +1
- Actual duration of study medication (Days) in cycle1 = sum of days with the administration of study
  medication during cycle 1, Dose interruption will be excluded from actual duration of exposure
- Actual duration of study medication (Days) for overall = sum of days with the administration of study medication, Dose interruption will be excluded from actual duration of exposure
- Cumulative dose of study medication (mg) in cycle 1 = Sum [Actual Daily Dose (mg/day) \* (Start Date of Administration – Stop Date of Administration + 1) of each record in cycle 1 in "Study Drug Administration" form. For patients who did not receive any dose of study medication, the cumulative dose will be set to zero
- Cumulative dose of study medication (mg) for overall = Sum [Actual Daily Dose (mg/day) \* (Start Date of Administration – Stop Date of Administration + 1) of each record in "Study Drug Administration" form.
   For patients who did not receive any dose of study medication, the cumulative dose will be set to zero
- Dose intensity (%) = Cumulative dose of study medication/ Total duration of study medication for each period (cycle 1 or overall)
- Relative dose intensity (%) = 100%\*Dose intensity/planned dose intensity, in this study, planned dose


intensity in each dose level is just the planned dose with unit of mg/day.

# 16. EFFICACY OUTCOMES

Efficacy data will be summarized by dose cohort in dose escalation phase and by disease cohort in dose expansion phase. PFS and OS will be analyzed for the SAS. The other efficacy variables (BOR, ORR, DCR, TTR, and DOR) will be analyzed for EAS.

Treatment efficacy will be evaluated by using tumor responses which will be assessed and documented at Screening, Day 1 of Cycle 2 and every 8 (+/-1 week) weeks on Day 1 of every other cycles afterwards (i.e. Cycle 4, 6... etc), until the occurrence of progressive disease (PD) according to the standard of Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Confirmation of CR and PR is required at no less than 4-week intervals between the date of initial response/progression and the confirmation assessment date. When the patient interrupts study medication due to AEs or other reasons, the evaluation should be conducted as scheduled. For suspected cases of PD before the start of the next scheduled assessment, additional tumor assessments will be done.

Tumor responses data are captured on CRF page "Tumor Measurement - Target Lesions", "Tumor Assessment - Non-Target lesions", "Tumor Assessment - New Lesions" and "Assessment of Disease". The confirmed best overall response (BOR, refer Section 16.1.2) will be summarized for EAS and will be presented together with summaries for objective response rate (ORR) and disease control rate (DCR).

The baseline sum of diameters will be presented with other baseline characteristics.

Tumor assessments for target lesion, non-target lesion, and new lesion will be presented in a listing. In addition, a listing of overall response including lesion responses, sum of diameters, and the corresponding change from baseline in tumor diameter will be provided.

Tumor assessment performed at the treatment completion visit (details can be found in SAP Section 7.3) is an eligible data point for the derivation of all efficacy endpoints, following the derivation rules described in Section 16.1.

## 16.1. EFFICACY VARIABLE(S) & DERIVATION(S)

#### 16.1.1. Progression-Free Survival

Progression-free survival (PFS) is defined as the time (in months) from the start date of study medication (Day 1) until the date of objective disease progression as defined by RECIST Version 1.1 or death (by any cause in the absence of progression), whichever occurred earlier.

The PFS time will always be derived based on scan/assessment dates and not based on visit dates. RECIST


assessments/scans contributing towards a particular visit, which consists of assessment for "Non-Target lesions", "Target lesions", and "New lesions", may be performed on different dates. The following rules will be applied:

- Date of progression will be determined based on the earliest of the dates of the radiological component that triggered the progression.
- When censoring a patient for PFS the patient will be censored at the latest of the dates contributing to a
  particular overall visit assessment.

If a patient has not experienced progressive disease (PD) or died before the end of study for any reason, progressionfree survival will be censored at the date of the last evaluable tumor assessment on or prior to the PD, which is not necessarily confirmed.

Three additional rules apply to PFS only:

- If a patient misses two or more consecutive tumor assessment visits, and showed PD or death afterwards, PFS will be censored at the date of last tumor assessment prior to the consecutive missed visits. Two consecutive missed/non-evaluable tumor assessment visit window is calculated as 2\*(8 weeks+1week window time), which is 126 days.
- If a patient reports no baseline tumor assessments or has no evaluable tumor assessment visits after the first
  dose of study medication, PFS will be censored at the start date of study medication unless they die within
  two consecutive tumor assessments since the first dose of study medication, i.e., PFS=1 day.
- Of note that tumor assessments after the first new anti-cancer treatment (same day inclusive) will be
  considered inadequate. If a patient starts new anti-tumor therapy initiated prior to documented disease
  progression or death on study, PFS will be censored at the date of the last tumor assessment prior to or on
  the date of new anti-tumor therapy.

See Table 1 for the detailed information of event/censoring rules for PFS:

Table 1: PFS Events/censoring rules

| Description | Event/Censor | Date of Event/Censor |
|---|---|---|
| Documented progression before start use of<br>new anti-tumor therapy and no two consecutive<br>missed tumor assessment visits | Event | Date of documented disease progression |
| Death without progression and without use of<br>new anti-tumor therapy and without missing<br>two consecutive tumor assessment visits | Event | Date of death |
| Death or progression after two or more consecutive missed tumor assessments | Censor | Date of last evaluable tumor assessment prior to the consecutive missed tumor |


| | | assessment visits |
|---|---|---|
| No evaluable baseline or post-baseline tumor<br>assessment and no new lesion found and no<br>death within two scheduled tumor assessment<br>visits post-baseline | Censor | Date of first dosing of study medication |
| New anti-tumor therapy started prior to<br>documented disease progression or death on<br>study | Censor | Date of last evaluable tumor assessment before start use of new anti-tumor therapy |
| No progression and no death before end of study or data cut-off | Censor | Date of last evaluable tumor assessment |

Note: Symptomatic deterioration will not be regarded as a progression event.

The PFS will be programmatically derived as follows:

- 1. If a patient had disease progression or death, then
- PFS (month) = ([date of earliest evidence of disease progression or death (including death from any cause) start date of study medication] + 1)/ 30.4375; Otherwise,
- 2. If the patient was known to have developed one of above censoring criteria, then the PFS is censored and PFS (month) = ([date of censoring start date of study medication] + 1)/ 30.4375.
- 3. Special scenario such as two or more consecutive missing tumor assessment visits or new anti-cancer treatment will be handled according to the rules provided in Table 1.

#### 16.1.2. Best Overall Response

Best overall response (BOR) will be calculated based on the overall visit responses obtained up until RECIST progression is documented, irrespective of whether patients discontinued study medication. In the absence of RECIST progression, BOR is determined by using visit responses up until the last evaluable overall visit response. Note, CR or PR response(s) after receiving subsequent anti-cancer therapy will not be included.

A patient's overall best objective response will be determined:

- CR: At least one visit response of CR confirmed by subsequent imaging at least 25 days (4 weeks 3 days window) later with no evidence of progression between confirmation visits. It is required that there is no other overall response, except CR and NE, between the first CR and the subsequent confirming CR which meet the confirmed CR criteria, i.e. CR-NE-CR is the confirmed CR.
- PR: At least one visit response of PR confirmed by subsequent imaging at least 25 days (4 weeks 3 days window) later with no evidence of progression between confirmation visits. It is required that there is no other overall response, except CR or PR or NE, between the first PR and the subsequent confirming CR or


PR which meet the confirmed CR or PR criteria, i.e PR-NE-PR is the confirmed PR. If the first PR followed by SD and no matter the requirement of SD is satisfied or not, i.e. PR-SD-PR, the subsequent PR will not be qualified as confirmed PR.

- SD needs to sustain for at least 8 weeks: Stable disease recorded at least 53 days after start of treatment (8 weeks from start of treatment, and also allowing a 3-day visit window). For example, an overall visit response of SD on day 28 will not be considered as SD.
- PD: Progression, or death in the absence of CR/PR or SD.
- NE: No evidence of CR/PR or SD or PD or death.
- Unconfirmed CR: If the BOR is not qualified as confirmed CR or PR but with at least one visit response of CR prior to subsequent new anti-tumor therapy or PD, then it will be considered as unconfirmed CR.
- Unconfirmed PR: If the BOR is not qualified as confirmed CR or PR but with at least one visit response of PR prior to subsequent new anti-tumor therapy or PD, then it will be considered as unconfirmed PR.

In addition, following special scenarios shall be considered for the determination of BOR:

 If a patient receives new anti-tumor therapy(s), for that patient, tumor assessments after the first new antitumor therapy (same day inclusive) will be considered inadequate, thus not counted towards the determination of BOR.

The table below illustrates the derivation of BOR (with confirmed response) and BOR (regardless of confirmation). Category of confirmed response is dependent on response at the subsequent time-point, and whether the minimum duration criterion for SD has been satisfied.

| Overall Response | Overall Response at | SD Sustaining | BOR Based on | BOR Regardless of |
|---|---|---|---|---|
| at First Time- | Subsequent Time- | Duration Met at | the Two Visits | Confirmation (for |
| point | point | First Time-point | | Unconfirmed CR or |
| | | | | PR) |
| CR | CR | Yes/No | CR | CR |
| CR | PR | Yes/No | SD/PD | CR (Unconfirmed) |
| CR | SD | Yes/No | SD/PD | CR (Unconfirmed) |
| CR | PD | Yes/No | SD/PD | CR (Unconfirmed) |


| CR | NE | Yes/No | SD/NE | CR (Unconfirmed) |
|----|----|--------|-------|------------------|
| PR | CR | Yes/No | PR/PR | PR |
| PR | PR | Yes/No | PR | PR |
| PR | SD | Yes/No | SD/SD | PR (Unconfirmed) |
| PR | PD | Yes/No | SD/PD | PR (Unconfirmed) |
| PR | NE | Yes/No | SD/NE | PR (Unconfirmed) |
| NE | NE | Yes/No | NE | NE |

CR = Complete Response; NE = Not Evaluable; ORR = Objective Response Rate; PD = Progressive Disease; PR= Partial Response; SD = Stable Disease.

For patients who progress and subsequently have a response, then the best objective response is only derived from assessments up to and including the time of the progression (i.e., it will not include the response after the patient has progressed).

Tumor response data for dosed patients that had non-measurable disease at baseline (i.e. did not meet study inclusion criteria 7) will be flagged and reviewed according to procedures described in Appendix 3 of the protocol.

#### 16.1.3. Objective Response Rate

Objective response rate (ORR) is defined as the proportion of patients with a best overall complete response (CR) or partial response (PR) per RECIST V.1.1. To be assigned a status of PR or CR, changes in tumor measurement must be confirmed by repeat assessment performed no less than 4 weeks after the criteria for response are first met. ORR (regardless of confirmation) will also be computed separately, including in the numerator subjects who have CR, unconfirmed CR, PR or unconfirmed PR. The denominator for the calculation of ORR and ORR regardless of confirmation will include all patients in EAS.

#### 16.1.4. Disease Control Rate

Disease control rate (DCR) is defined as the proportion of patients whose best overall response from baseline is either CR, PR, or SD per RECIST v.1.1. The denominator for the calculation of DCR will include all patients in EAS subset of response evaluable patients. Response evaluable patients refer to patients with a baseline RECIST assessment.


### 16.1.5. Time to Response

Time to response (TTR) is defined as the time between the start date of study medication until first documented response (CR or PR, which is subsequently confirmed) according to RECIST v.1.1. Time to response is only applicable to patients whose BOR is either CR or PR. TTR (months) will be calculated as (First CR/PR date – start date of study medication + 1) / 30.4375.

### 16.1.6. Duration of Objective Response

Duration of objective response (DoR) is defined as the time from the first time that the objective response reaches CR or PR, whichever comes first, until the occurrence of PD or death (if the death of the patient occurs before recording the PD). If the response is not confirmed, it will not be included. If a patient does not progress (or does not progress before receiving new anti-cancer treatment) following a response, then their duration of response will use the PFS censoring time.

For those patients with confirmed response, the date of response will be the date of first documented response, not the date of confirmatory tumor assessment for that response. The DoR (months) will be calculated as (PD/Death date - First CR/PR date + 1) / 30.4375 when a patient is deemed to experience a PFS event after first CR/PR, or calculated as (PFS censoring date - First CR/PR date +1)/30.4375 when a patient is deemed to be censored.

#### 16.1.7. Percentage Change in Tumor Size

Percentage change in tumor size will be determined for patients with measurable disease at baseline and is derived at each visit by the percentage change in the sum of the diameters of target lesions compared to baseline. Best (minimum) percentage change from baseline (PCFB) in tumor size will be summarized by dose cohort and disease cohort using descriptive statistics and a waterfall plot will be presented also. The sum of diameters will be taken from the field "Sum of Diameters of Target Lesions" in "Assessment of Disease (According to RECIST 1.1) (RS)" form of eCRF or be calculated from the field "Measured Diameter" in "Tumor Results: Target Lesion (TARGET)" form of eCRF.

#### 16.2. PRIMARY ANALYSIS OF EFFICACY VARIABLE(S)

For each dose level in dose escalation phase and each disease cohort in dose expansion phase, PFS will be described in tabular and graphical format using Kaplan-Meier methods, including estimated median (in months) with 95% CI, 25th and 75th percentiles, minimum, maximum. The 95% CI for the median survival time will be derived using the log-log transformation based on Brookmeyer and Crowley method.

Besides, Kaplan-Meier estimated probabilities with corresponding 80% and 95% CIs at several time points


(including 4 Months/ 16 Weeks and 11 months) will also be provided and the 80% and 95% CIs will be derived using the log-log transformation based on Greenwood's formula.

Censoring reasons will also be summarized by categories that will be determined using the treatment completion page, the study evaluation completion page and survival page.

The other endpoints including TTR and DoR will be analyzed in the same way where appropriate. In case the number of responses in each treatment group is very small, DoR and TTR may be listed only.

ORR and DCR will be estimated and 95% exact confidence intervals (CIs) based on the Clopper-Pearson method will be presented.

The time to event/censoring and the censoring status for PFS will be listed for the SAS, and for DOR and BOR will be listed for the EAS.

#### 16.3. EXPLORATORY EFFICACY

#### 16.3.1. Tumor Markers

Tumor markers may include, but are not limited to, serum CEA and CA 19-9 (patients with BTC) serum chromogranin A (CgA) and neuron-specific enolase (NSE) for patients with pNET and epNET; and serum or plasma VEGF for all diseases cohorts. Assessment of tumor markers will be performed within 28 days prior to the start of treatment with study drug (C1D1) and at each tumor assessment visit.

The values and change from baseline in tumor markers will be summarized by disease cohort (BTC, pNET, or epNET, or STS) using descriptive statistics. The individual tumor marker test results will be listed by dose cohorts in each phase and by patients. Other exploratory analyses may be performed as appropriate.

#### 16.3.2. Overall Survival

Overall survival (OS) (in months) is defined as the time interval between the start date of study drug and the date of patient death (any cause). The final known date alive will be used as the censoring date for patients who have not been reported to have died by the time of analysis cut-off date. OS will be analyzed for only the BTC and STS cohorts based on the SAS.

Patients who fail to provide any follow-up information will be censored on the date of enrolment. OS (months) will be calculated as (Date of death – start date of study medication + 1) / 30.4375.


Median, 25<sup>th</sup> and 75<sup>th</sup> Quartiles, minimum and maximum will be provided for OS. Kaplan-Meier estimated probabilities with corresponding 80% and 95% CIs at several time points (including 16 weeks, 6 months, 8 months and 11 months for BTC and STS cohort) will be provided. Kaplan-Meier curves will be constructed to provide a visual presentation of the OS change with time.

### 16.4. SENSITIVITY ANALYSIS OF EFFICACY VARIABLE(S)

No sensitivity or supportive analyses will be performed on efficacy variables.

# 17. SAFETY OUTCOMES

All outputs for safety outcomes except DLT summary will be based on the SAS. Safety data will be summarized by dose cohort in escalation phase and disease cohort in dose expansion phase.

#### 17.1. ADVERSE EVENTS

An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the investigational medicinal product or other protocol-imposed intervention, regardless of attribution.

Relevant information is recorded on CRF page "Adverse Event/Serious Adverse Event".

If a persistent AE becomes more severe, it should be recorded again with the updated severity. All recurrent AEs (AEs that occurs and resolves between patient evaluation time points and subsequently recurs) should be recorded on "Adverse Event/Serious Adverse Event" CRF.

A pre-existing medical condition should be recorded as an AE or SAE only if the frequency, severity, or character of the condition worsens during the study.

After informed consent, but prior to initiation of study medications, only SAEs caused by a protocol-mandated intervention will be collected.

After initiation of study medications, all AEs and SAEs regardless of attribution will be collected until 37 days (30 days + 7 days window) following the last administration of study medication or study discontinuation/termination, whichever is later. After this period, investigators should report only SAEs that are felt to be related to prior study treatment.

Treatment-emergent AEs (TEAEs) are defined as AEs that started or worsened in severity on or after the first administration date of study medication and no later than 30 (+7) days after the last administration date of study


medication or initiation of new anti-tumor therapy (whichever occurs first).

An exception is that study medication related SAEs collected later than 37 days after the last dosing date will be treated as TEAEs.

If the start date coincides with the reference start date, a query "Prior/ post 1st dose" will be used to identify TEAEs (only when 'Post 1st dose' will be considered as TEAE, if 'Prior' then not TEAE). When there is no definite answer to the query, the AE will be considered as a TEAE. See section 8.2 for handling of partial dates for AEs. In the case where it is not possible to classify an AE as treatment-emergent or not, the AE will be classified by the worst case; i.e. treatment-emergent.

If a subject reports a TEAE more than once in the SOC/PT, the TEAE with highest severity will be used in the corresponding summaries.

An overall summary of number of patients within each of the categories described in the sub-section below, will be provided for all AEs as specified in the templates.

For all SOC/PT summaries, AEs will be presented in alphabetic order except the uncoded SOC/PT. Uncoded SOC/PT will be presented as "Uncoded" and be presented at the end of relevant AE summaries.

A Listing of all AEs with relevant information being reported during study with flag to distinguish TEAE and Non-TEAE will be provided.

#### 17.1.1. All TEAEs

In the analysis of AEs, the MedDRA adverse event dictionary Version 23.0 or higher will be used to map verbatim terms to SOC and PT.

An overall summary of TEAEs including severity, relationship, action taken, and outcome will be provided. Incidence of TEAEs will be presented by SOC and then PT and also broken down further by maximum severity (Section 17.1.1.1) and relationship to study medication (Section 17.1.1.2) for each dose level, and each disease cohort. Number (n) and percentage (%) will be presented with the % calculated relative to the total number of patients in the SAS. In the case that a patient report multiple TEAEs, the TEAE with worst severity and strongest relationship (related to study medication) will be used in the corresponding summaries.

### 17.1.1.1 Severity

The severity of all TEAEs will be graded according to 5 grades (Grade 1 to Grade 5) in accordance with the National Cancer Institute Common Terminology criteria for adverse events (NCI-CTCAE) V4.03 as defined in the Study Protocol Section 7.1.5.

TEAEs missing severity will be classified as Grade 3.

TEAEs of each severity grade will be summarized using incidence (frequencies and percentages) by SOC and PT will be summarized by dose level in the dose escalation phase and by disease cohort in the dose expansion phase. If


a patient reports a TEAE more than once within that SOC/ PT, the AE with the worst case severity will be used in the corresponding severity summaries.

### 17.1.1.2 Relationship to Study Medication

As indicated by the Investigator, causal relationship between AEs and study medication will be classified as "reasonably possible" or not. TEAEs with missing relationship to study medication will be regarded related. Related and Not Related TEAEs will be summarized by dose level in dose escalation phase, and by disease cohort in dose expansion phase using incidence (frequencies and percentages) by SOC and PT. If a patient reports the same AE more than once within that SOC/PT, the AE with the worst relationship (ie, related) to study medication will be used in the corresponding relationship summaries.

### 17.1.2. TEAEs Leading to Discontinuation of Study Medication

TEAEs leading to permanent discontinuation of study medication will be identified as those records with a response of "Drug Withdrawn" to the item "Action taken with the study drug" on the "Adverse Event/Serious Adverse Event (AE/SAE)" form of the CRF.

For TEAEs leading to drug discontinuation, summaries of incidence (frequencies and percentages) by SOC and PT will be prepared. Summaries for TEAEs leading to discontinuation of study medication by SOC and PT will be further broken down by maximum severity and relationship to study medication.

#### 17.1.3. TEAEs Leading to Study Medication Adjustment

TEAEs leading to study medication adjustment will be identified as those records with a response of "Drug interrupted" or "Dose reduced" or 'Dose increased' to the item "Action taken with the study drug" on the AE/SAE form of the CRF.

For TEAEs leading to study medication adjustment, summaries of incidence (frequencies and percentages) by SOC and PT will be prepared. Summaries for TEAEs leading to study medication adjustment by SOC and PT will be further broken down by maximum severity and strongest relationship to study medication.

#### 17.1.4. Serious TEAEs

A serious adverse event (SAE) is defined as any life-threatening AE resulting in death, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or any other important medical event requiring intervention, in-patient hospitalization or prolongation of existing hospitalization.

Detailed definition of SAEs can be found in Protocol Section 9.1.1.

On the CRF, SAEs are those events with a response of "Yes" for the item "Does the Adverse Event meet seriousness criteria?". Summaries of incidence (frequencies and percentages) of serious TEAEs by SOC and PT will be


prepared. In addition, summaries for serious TEAEs by SOC and PT will be further broken down by maximum severity and strongest relationship to study medication.

SAEs will be flagged and included in a listing of AEs.

### 17.1.5. TEAEs Of Special Interest (TEAESI)

The preferred terms for TEAESI are included in Appendix 2. Summaries of incidence (frequencies and percentages) of TEAESIs by Standardized MedDRA Queries (SMQ) and PT based on the <a href="Appendix 2">Appendix 2</a> will be prepared. The broad search will be used for SMQ terms. Time to TEAESI onset is defined as time interval from date of first administration of study medication to the earliest onset date among TEAEs within the same SMQ. Time to TEAESI onset will be summarized by SMQ for each dose cohort and disease cohort.

AESIs will be flagged and included in a listing of AEs.

### 17.1.6. Dose Limiting Toxicity (DLT)

A detailed definition of DLT can be found in Protocol Section 4.1.2. On the CRF, DLT will be identified among all AEs using question "Is it DLT?", and details will be captured on CRF page "DLT Assessment". Incidence of DLTs by SOC and PT will be summarized for DLT set. Time between date of first dose of study medication and DLT event onset will be presented for DLT evaluable set.

All relevant information of DLT assessment will be listed for DLT evaluable set by dose cohort and by patient.

#### 17.1.7. Deaths

If any patients die during the study conduct, as recorded on the "Death" CRF form, the count and cause of death and on treatment death (event occurs on or after first study medication dose and prior to 37 days [30 days + 7 days window] after the last dose) will be summarized by dose level in dose escalation phase, and by disease cohort in dose expansion phase.

Individual information of subject ID, death date and primary reason for death will be presented in the listing. Ontreatment death will be flagged.

### 17.2. LABORATORY EVALUATIONS

Laboratory samples will be analyzed at the study site's local laboratory. Laboratory assessments will include the following:

- Hematology, which is recorded on CRF page "LAB Hematology"
- Coagulation, INR and aPTT, which is captured on CRF page "LAB Coagulation".


- Serum chemistry, which is recorded on CRF page "LAB Blood Chemistry"
- Serum pregnancy test at screening for all women of childbearing potential, which is captured on CRF page "Pregnancy Test"
- Urinalysis, which is recorded on CRF page "LAB Urinalysis" and "LAB-24hrs Urine Protein"
- Thyroid function: TSH, free T3, free T4, which is captured on CRF page "LAB Thyroid Function Tests"
- Stool occult blood test, which is recorded on CRF page "LAB Fecal Occult Blood Test"

Test normal ranges of all quantitative tests above (ie, all tests excluding stool occult blood test and serum pregnancy test) are also recorded on corresponding normal range CRF pages.

Data recorded by the laboratory will be converted to the International System of Units (SI) and all presentations will use SI units. Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of normal range (LLN), or "> X", i.e. above the upper limit of normal range (ULN), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

The following summaries will be provided for laboratory data:

- For quantitative results, actual value of each scheduled visit, change from baseline for each post-baseline scheduled measurement.
- For quantitative measurements and categorical measurements, Incidence of abnormal values assessed by investigator. Shift from baseline according to markedly abnormal criteria based on investigators' assessment.
- Shift from baseline to worst grade in CTCAE grade according to Common Toxicity (CTC) grading system for parameters of hematology and serum biochemistry whose CTCAE scale is available.
- Listing of all laboratory data by patient, abnormal values identified according to normal range (low, normal
  and high), and markedly abnormal criteria by investigators' assessment will be flagged.

#### 17.2.1. Laboratory Specific Derivations

Creatinine clearance (CCr) will be calculated by using the serum creatinine (SCr) values according to the the following formulas:

- Male: CCr = [(140 age) × weight (kg)] / [0.818 × SCr (umol/L)]
- Female: CCr = [(140 age) × weight (kg)] / [0.818 × SCr (umol/L)] × 0.85

The units for creatinine clearance will be converted to SI unit: umol/L.

# 17.2.2. Laboratory Reference Ranges and Markedly Abnormal Criteria

All laboratory assessments except serum pregnancy test and stool occult blood test will be analyzed as following.

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and


categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

In addition to the high and low quantitative laboratory assignments (as identified by means of the laboratory reference ranges), markedly abnormal quantitative safety (and other) laboratory assessments will also be evaluated as normal/abnormal, not clinically significant (NCS)/ abnormal, clinically significant (CS) by investigator. For laboratory assessments collected with both quantitative and qualitative results, if most assessments are quantitative, quantitative assessments will be summarized, and vice versa if most assessments are qualitative, and all the assessments will be listed.

# 17.2.3. CTCAE Grading for Laboratory Data

Quantitative laboratory measurements will be graded according to NCI CTCAE V4.03 wherever applicable. All grading will be based on lab values (being direct or some derived, corrected values) ONLY, regardless of its interventional or symptomatic consequences.

Some modifications to the grading system will be applied:

- Grade 5 refers to fatal outcomes, which cannot be determined solely by lab values, therefore will not appear
  in the grading system. In addition to the usual defined categories.
- A further category denoted Grade 0 will include all other laboratory values except missing values.
- Missing results shall be graded as missing.

For some specific parameters with CTCAE grading in both high and low direction (e.g., calcium, glucose, magnesium, potassium, sodium), CTCAE in high and low directions will be presented separately, i.e. hyper for higher values of concern and hypo for lower values of concern.

Shifts in toxicity grade from baseline to the worst toxicity grade will be provided for the SAS.

#### 17.2.4. Liver Function Abnormality

Liver function abnormality is defined in Protocol Section 7.1.7 and the below events will be identified via programming and summarized by categories and dose cohort for SAS. Separate listings for patients with drug-induced liver injury (DILI) will also be provided.

- ALT/AST > 3 x ULN and ≤ 5 x ULN
- ALT/AST > 5 x ULN
- Total Bilirubin > 2 x ULN
- ALT/AST > 3 x ULN AND concurrent Total bilirubin > 2 x ULN


#### 17.3. ECG EVALUATIONS

The 12- Lead Electrocardiogram (ECG) will be performed at screening, and on Days 1 and 15 in Cycle 1. when ECG data will be collected at pre-dose and at 2 hours +-15 minutes post-dose (around C<sub>max</sub> after single dose and at steady state in order to evaluate concentration-QT relationship for surufatinib). The ECG values at C1D1 pre-dose will be used as 'baseline' value in the analysis. ECG will also be conducted on Day 1 of each cycle from Cycle 2 and onward, as well as the treatment completion visit.

For each time-point, following measurements with change from baseline values will be presented for the SAS:

- Heart rate (bpm)
- RR (ms)
- PR (ms)
- QRS (ms)
- QT (ms)
- QT correction by Bazett (ms)
- QT correction by Fridericia (ms)
- Overall ECG interpretation
  - Abnormal, clinically significant (CS)
  - Abnormal, not clinically significant (NCS)
  - Normal
  - Incomplete analysis
  - Uninterpretable
  - Not applicable

### 17.3.1. ECG Specific Derivations

There will be no specific derivations for ECG.

### 17.3.2. ECG Markedly Abnormal Criteria

The number and percentage of patients with notable ECG values at baseline and post-baseline will be summarized. These summaries will be done for worst post-baseline value for each category. The criteria for notable ECG values are provided in Table 2 below.

| Table 2 | Notab | le EC | G V | /alues |
|---------|-------|-------|-----|--------|

| Test | Notable ECG Values |
|------|--------------------|
|------|--------------------|




| QTcF/QTcB<br>(absolute) | interval >450 to 480 msec<br>interval >480 to 500 msec<br>interval >500 msec |
|---|---|
| Heart rate<br>(absolute) | <50 bpm<br>>100 bpm |
| PR (absolute) | interval >200 msec |
| QRS (absolute) | interval >120 msec |

#### •

# 17.3.3. Analysis of QTc Change from Baseline (ΔQTc)

The change from baseline in QTcF (ΔQTcF) intervals will be evaluated as follows:

- ΔQTcF at each time point will be listed for each patient and treatment. For each time point of measurement, ΔQTcF will be summarized using descriptive statistics (mean, SD, median, min, max).
- The incidence of patients with ΔQTcF increase >30 to 60 msec and >60 msec will be summarized.
- The incidence of patients with ΔQTcF increase >30 to 60 msec and >60 msec by time-point in Cycle 1 will also be summarized.
- Patients with ΔQTcF increase >60 msec will be listed.
- Mean ΔQTcF versus time profile for each dose group will be plotted on the same graph.

### 17.3.4. Analysis of the Relationship Between QT/QTc and RR at Baseline

The relationship between QT/QTc and RR intervals at baseline will be evaluated graphically as follows:

- The logarithm of baseline QT values will be plotted against the logarithm of corresponding RR intervals
- A linear regression model will be fitted to the data with logarithm of baseline QTc interval values as
  the dependent variable and logarithm of RR as the predictor.
- The slope of the regression line and its standard error, along with 2-sided 95% confidence intervals for the slope, will be estimated from this model.
- The analysis will be repeated for QTcB and QTcF and plotted on the same graph for QT.


# 17.4. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Systolic blood pressure (mmHg)
- Diastolic blood pressure (mmHg)
- Heart rate (beats/min)
- Respiratory Rate (breaths/min)
- Temperature (°C)
- Weight (kg)
- Baseline BMI (kg/m²)
- Baseline Height (cm)

Vital sign values and change from baseline (applicable to post-baseline measurements) will be summarized by each scheduled time-point.

All vital signs results including change from baseline for quantitative parameters will be listed. A flag of oral temperature derived from axillary temperature will be provided.

Selected vital signs (SBP, DBP and heart rate) change from baseline will be plotted over time for each patient.

# 17.4.1. Vital Signs Specific Derivations

There will be no specific derivations for vital signs.

### 17.4.2. Vital Signs Markedly Abnormal Criteria

Markedly abnormal quantitative Vital Signs measurements will be identified in accordance with the following predefined markedly abnormal criteria:

Table 3 Vital Sign Markedly Abnormal Criteria.

| Variable | Unit | Baseline | High |
|---|---|---|---|
| | | Category | |
| SBP | mmHg | ≤ 140 mmHg | Absolute change from baseline of:<br>> 0 - $\leq$ 20 / > 20 - $\leq$ 40 / > 40 mmHg |
| DBP | mmHg | ≤ 90 mmHg | Absolute change from baseline of: $> 0 - \le 20 / > 20 - \le 40 / > 40 \text{ mmHg}$ |


| Variable | Unit | Baseline | High |
|---|---|---|---|
| | | Category | |
| Heart rate | Bpm | < 100 / ≥ 100<br>bpm | Absolute change from baseline of: $> 0 - \le 20 / > 20 - \le 40 / > 40$ bpm |
| Weight | Kg | None | Percentage change from baseline of < 5% / $\geq$ 5 - <10% / $\geq$ 10 - < 20% / $\geq$ 20% |

#### 17.5. Physical Examination

A complete physical examination at screening should include the evaluation of head, eye, ear, nose, and throat; and cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, and neurological systems.

At subsequent visits, a limited physical examination will be performed to assess changes from baseline

At subsequent visits, a limited physical examination will be performed to assess changes from baseline abnormalities, any new abnormalities, and to evaluate patient-reported symptoms. New or worsened abnormalities should be recorded as AEs if appropriate.

All physical examination results will be listed.

#### 17.6. OTHER SAFETY ASSESSMENTS

#### 17.6.1. ECOG Performance Status

The Eastern Cooperative Oncology Group (ECOG) Performance Status will be summarized descriptively by visit and a shift table will be also summarized from the "ECOG Performance Status" CRF page. In addition, the summary descriptive table by visit will include specific ECOG grades and binary grouping grades (0-1, 2-5). The shift table will be summarized from baseline to worst post-baseline.

Details about ECOG performance status scores can be found in Protocol Appendix B.

A listing of ECOG Performance Status will be provided.

### 17.6.2. Echocardiogram

Echocardiography, including left ventricular ejection fraction (LVEF) assessment contains both quantitative results (%) and overall evaluation [Normal, Abnormal, Not Clinically Significant (ANCS); Abnormal, Clinically Significant (ACS)].

Actual value of echocardiography measured at each scheduled visit, change from baseline to each post-baseline




scheduled measurement will be presented by visit. Overall evaluation will be summarized separately.

All echocardiography results including change from baseline for LVEF and relevant information will be listed.

# 18. REFERENCES

Protocol 2015-012-00US1 Version 7.0 (Amendment 11), Dated 19Mar2021 Case Report Forms Version 11 Dated 30Aug2021


# APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

# **IQVIA OUTPUT CONVENTIONS**

Outputs will be presented according to the Quintiles' general guidelines and template for outputs conventions.

# **DATES & TIMES**

Depending on data available, dates and times will take the form DDMMMYYYY and HH:MM:SS.

# SPELLING FORMAT

English US.

# PRESENTATION OF TREATMENT GROUPS

All summaries will be presented by assigned dose level in dose escalation phase.

| Treatment Group | For Tables, Listings and Graphs |
|---|---|
| 50 mg/day dose level | 50 mg |
| 100 mg/day dose level | 100 mg |
| 200 mg/day dose level | 200 mg |
| 300 mg/day dose level | 300 mg |
| 400 mg/day dose level | 400 mg |
| Additional intermediate dose level | XXX mg (XXX=Actual dose level) |
| Screen failures (in listings only) | SF |
| Untreated eligible patients (in listings only) | NOTTRT |


# PRESENTATION OF DISEASE COHORT

All summaries will be presented by disease cohort in dose expansion phase.

| Disease Cohort | For Tables, Listings and Graphs |
|---|---|
| Arm A: Biliary tract cancer | BTC |
| Arm B: Pancreatic neuroendocrine tumor | pNET |
| Arm C: Extrapancreatic neuroendocrine tumor | epNET |
| Arm D: Soft tissue sarcoma | STS |

# PRESENTING ORDER

All listings will be ordered by the following (unless otherwise indicated in the template):

- SitePatient ID,
- · Treatment group, in the order as above table,
- date (where applicable)

All tables containing coded terms (CM, MH, AE, etc), coded records will be sorted in descending order of incidence.

# APPENDIX 2. ADVERSE EVENTS OF SPECIAL INTEREST

| AESI SMQ | PT Term | PT Code |
|-------------|-------------------------------|----------|
| Acute renal | Acute kidney injury | 10069339 |
| failure | Acute phosphate nephropathy | 10069688 |
| | Anuria | 10002847 |
| | Azotaemia | 10003885 |
| | Continuous haemodiafiltration | 10066338 |
| | Dialysis | 10061105 |
| | Foetal renal impairment | 10078987 |
| | Haemodialysis | 10018875 |
| | Haemofiltration | 10053090 |




| | Neonatal anuria | 10049778 |
|--------------|---------------------------------------------------|----------|
| | Nephropathy toxic | 10029155 |
| | Oliguria | 10030302 |
| | Peritoneal dialysis | 10034660 |
| | Prerenal failure | 10072370 |
| | Renal failure | 10038435 |
| | Renal failure neonatal | 10038447 |
| | Renal impairment | 10062237 |
| | Renal impairment neonatal | 10049776 |
| | Subacute kidney injury | 10081980 |
| Haemorrhages | Abdominal wall haematoma | 10067383 |
| | Abdominal wall haemorrhage | 10067788 |
| | Abnormal withdrawal bleeding | 10069195 |
| | Achenbach syndrome | 10079562 |
| | Acute haemorrhagic leukoencephalitis | 10058994 |
| | Acute haemorrhagic ulcerative colitis | 10075634 |
| | Administration site bruise | 10075094 |
| | Administration site baematoma | 10075100 |
| | | 10075100 |
| | Administration site haemorrhage Adrenal haematoma | |
| | Total International | 10059194 |
| | Adrenal haemorrhage | 10001361 |
| | Anal fissure haemorrhage | 10079765 |
| | Anal haemorrhage | 10049555 |
| | Anal ulcer haemorrhage | 10063896 |
| | Anastomotic haemorrhage | 10056346 |
| | Anastomotic ulcer haemorrhage | 10002244 |
| | Aneurysm ruptured | 10048380 |
| | Angina bullosa haemorrhagica | 10064223 |
| | Anorectal varices haemorrhage | 10068925 |
| | Anticoagulant-related nephropathy | 10083346 |
| | Aortic aneurysm rupture | 10002886 |
| | Aortic dissection rupture | 10068119 |
| | Aortic intramural haematoma | 10067975 |
| | Aortic perforation | 10075729 |
| | Aortic rupture | 10060874 |
| | Aponeurosis contusion | 10075330 |
| | Application site bruise | 10050114 |
| | Application site haematoma | 10068317 |
| | Application site haemorrhage | 10072694 |
| | Application site purpura | 10072094 |
| | Arterial haemorrhage | 10050182 |
| | Arterial intramural haematoma | |
| | | 10074971 |
| | Arterial perforation | 10075732 |
| | Arterial rupture | 10003173 |
| | Arteriovenous fistula site haematoma | 10055150 |
| | Arteriovenous fistula site haemorrhage | 10055123 |
| | Arteriovenous graft site haematoma | 10055152 |




| Arteriovenous graft site haemorrhage | 10055126 |
|--------------------------------------------------|----------|
| | I . |
| Astringent therapy | 10067372 |
| Atrial rupture | 10048761 |
| Auricular haematoma | 10003797 |
| Basal ganglia haematoma | 10077031 |
| Basal ganglia haemorrhage | 10067057 |
| Basilar artery perforation | 10075736 |
| Bladder tamponade | 10062656 |
| Bleeding varicose vein | 10005144 |
| Blood blister | 10005372 |
| Blood loss anaemia | 10082297 |
| Blood urine | 10005863 |
| Blood urine present | 10018870 |
| Bloody discharge | 10057687 |
| Bloody peritoneal effluent | 10067442 |
| Bone contusion | 10066251 |
| Bone marrow haemorrhage | 10073581 |
| Brain confusion | 10052346 |
| Brain stem haematoma | 10073230 |
| Brain stem haemorrhage | 10006145 |
| Brain stem microhaemorrhage | 10071205 |
| Breast haematoma | 10064753 |
| Breast haemorrhage | 10004755 |
| Broad ligament haematoma | 10006254 |
| Bronchial haemorrhage | 10065739 |
| Bronchial varices haemorrhage | 10079163 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Bursal haematoma | 10077818 |
| Cardiac contusion | 10073356 |
| Carotid aneurysm rupture | 10051328 |
| Carotid artery perforation | 10075728 |
| Catheter site bruise | 10063587 |
| Catheter site haematoma | 10055662 |
| Catheter site haemorrhage | 10051099 |
| Central nervous system haemorrhage | 10072043 |
| Cephalhaematoma | 10008014 |
| Cerebellar haematoma | 10061038 |
| Cerebellar haemorrhage | 10008030 |
| Cerebellar microhaemorrhage | 10071206 |
| Cerebral aneurysm perforation | 10075394 |
| Cerebral aneurysm ruptured syphilitic | 10008076 |
| Cerebral arteriovenous malformation haemorrhagic | 10008086 |
| Cerebral artery perforation | 10075734 |
| Cerebral cyst haemorrhage | 10082099 |
| Cerebral haematoma | 10053942 |
| Cerebral haemorrhage | 10008111 |
| Cerebral haemorrhage foetal | 10050111 |
| Colora nacinomage rocar | 10030137 |




| Cerebral haemorrhage neonatal | 10008112 |
|---------------------------------------|----------|
| 8 | 10067277 |
| | 10050020 |
| 8 | 10050022 |
| | 10076597 |
| | 10068642 |
| 8 | 10008786 |
| | 10050399 |
| | 10072726 |
| | 10057417 |
| | 10065019 |
| | 10009996 |
| | 10010719 |
| | 10050584 |
| Comeal bleeding | 10051558 |
| Cullen's sign | 10059029 |
| Cystitis haemorrhagic | 10011793 |
| Deep dissecting haematoma | 10074718 |
| Diarrhoea haemorrhagic | 10012741 |
| _ | 10013442 |
| | 10013541 |
| | 10013560 |
| | 10013839 |
| 8 | 10013865 |
| | 10013908 |
| | 10014009 |
| | 10014080 |
| | 10014589 |
| | 10014896 |
| | 10073681 |
| | 10015090 |
| | 10015719 |
| | 10078254 |
| · | |
| | 10015769 |
| | 10082797 |
| | 10015867 |
| | 10073354 |
| — j | 10079891 |
| | 10015926 |
| , , | 10053196 |
| | 10075018 |
| | 10064976 |
| | 10075739 |
| | 10075745 |
| | 10016871 |
| | 10081749 |
| Gastric haemorrhage | 10017788 |




| Gastric ulcer haemorrhage | 10017826 |
|-----------------------------------------------------|----------|
| Gastric ulcer haemorrhage, obstructive | 10017829 |
| Gastric varices haemorrhage | 10057572 |
| Gastritis alcoholic haemorrhagic | 10017857 |
| Gastritis haemorrhagic | 10017866 |
| Gastroduodenal haemorrhage | 10053768 |
| Gastrointestinal haemorrhage | 10017955 |
| Gastrointestinal polyp haemorrhage | 10074437 |
| Gastrointestinal ulcer haemorrhage | 10056743 |
| Gastrointestinal vascular malformation haemorrhagic | 10080561 |
| Genital contusion | 10073355 |
| Genital haemorrhage | 10061178 |
| Gingival bleeding | 10018276 |
| Graft haemorrhage | 10063577 |
| Grey Turner's sign | 10075426 |
| Haemangioma rupture | 10084040 |
| Haemarthrosis | 10018829 |
| Haematemesis | 10018830 |
| Haematochezia | 10018836 |
| Haematocoele | 10018833 |
| Haematoma | 10018852 |
| Haematoma evacuation | 10060733 |
| Haematoma infection | 10051564 |
| Haematoma muscle | 10055890 |
| Haematosalpinx | 10050468 |
| Haematospermia | 10018866 |
| Haematotympanum | 10063013 |
| Haematuria | 10018867 |
| Haematuria traumatic | 10018871 |
| Haemobilia | 10058947 |
| Haemoperitoneum | 10018935 |
| Haemophilic arthropathy | 10065057 |
| Haemophilic pseudotumour | 10073770 |
| Haemoptysis | 10018964 |
| Haemorrhage | 10055798 |
| Haemorrhage coronary artery | 10055803 |
| Haemorrhage foetal | 10061191 |
| Haemorrhage in pregnancy | 10018981 |
| Haemorrhage intracranial | 10018985 |
| Haemorrhage neonatal | 10061993 |
| Haemorrhage subcutaneous | 10018999 |
| Haemorrhage subepidermal | 10019001 |
| Haemorrhage urinary tract | 10055847 |
| Haemorrhagic adrenal infarction | 10079902 |
| Haemorrhagic arteriovenous malformation | 10064595 |
| Haemorrhagic ascites | 10059766 |
| Haemorrhagic breast cyst | 10077443 |




| | 4004000 |
|----------------------------------------|----------|
| Haemorrhagic cerebral infarction | 10019005 |
| Haemorrhagic cyst | 10059189 |
| Haemorrhagic diathesis | 10062713 |
| Haemorrhagic disease of newborn | 10019008 |
| Haemorrhagic disorder | 10019009 |
| Haemorrhagic erosive gastritis | 10067786 |
| Haemorrhagic hepatic cyst | 10067796 |
| Haemorrhagic infarction | 10019013 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Haemorrhagic ovarian cyst | 10060781 |
| Haemorrhagic stroke | 10000781 |
| Haemorrhagic thyroid cyst | 10072256 |
| Haemorrhagic transformation stroke | 10055677 |
| Haemorrhagic tumour necrosis | 10054096 |
| Haemorrhagic urticaria | 10059499 |
| Haemorrhagic vasculitis | 10071252 |
| Haemorrhoidal haemorrhage | 10054787 |
| Haemostasis | 10067439 |
| Haemothorax | 10019027 |
| Henoch-Schonlein purpura | 10019617 |
| Hepatic haemangioma rupture | 10054885 |
| Hepatic haematoma | 10019676 |
| Hepatic haemorrhage | 10019677 |
| Hereditary haemorrhagic telangiectasia | 10019883 |
| Hyperfibrinolysis | 10074737 |
| Hyphaema | 10020923 |
| Iliac artery perforation | 10075731 |
| Iliac artery rupture | 10072789 |
| Iliac vein perforation | 10072769 |
| Immune thrombocytopenia | 10073744 |
| Implant site bruising | 10063842 |
| Implant site haematoma | 10063780 |
| Implant site haemorrhage | 10053995 |
| Incision site haematoma | 10059241 |
| Incision site haemorrhage | 10051100 |
| Increased tendency to bruise | 10021688 |
| Induced abortion haemorrhage | 10052844 |
| Inferior vena cava perforation | 10075742 |
| Infusion site bruising | 10059203 |
| Infusion site haematoma | 10065463 |
| Infusion site haemorrhage | 10065464 |
| Injection site bruising | 10022052 |
| Injection site haematoma | 10022066 |
| Injection site haemorrhage | 10022067 |
| Instillation site bruise | 10073630 |
| Instillation site haematoma | 10073609 |
| Instillation site haemorrhage | 10073610 |
| AND HANDER OF THE PARTY HERE | 100/3010 |




| 7 . 44 | 10075100 |
|---------------------------------------|----------|
| Internal haemorrhage | 10075192 |
| Intestinal haematoma | 10069829 |
| Intestinal haemorrhage | 10059175 |
| Intestinal varices haemorrhage | 10078058 |
| Intra-abdominal haematoma | 10056457 |
| Intra-abdominal haemorrhage | 10061249 |
| Intracerebral haematoma evacuation | 10062025 |
| Intracranial haematoma | 10059491 |
| | 10039491 |
| Intracranial tumour haemorrhage | |
| Intraocular haematoma | 10071934 |
| Intrapartum haemorrhage | 10067703 |
| Intraventricular haemorrhage | 10022840 |
| Intraventricular haemorrhage neonatal | 10022841 |
| Iris haemorrhage | 10057418 |
| Joint microhaemorrhage | 10077666 |
| Kidney contusion | 10023413 |
| Lacrimal haemorrhage | 10069930 |
| Large intestinal haemorrhage | 10052534 |
| Large intestinal ulcer haemorrhage | 10061262 |
| Laryngeal haematoma | 10070885 |
| Laryngeal haemorrhage | 10070383 |
| , . | 10066304 |
| Lip haematoma | |
| Lip haemorrhage | 10049297 |
| Liver contusion | 10067266 |
| Lower gastrointestinal haemorrhage | 10050953 |
| Lower limb artery perforation | 10075730 |
| Lymph node haemorrhage | 10074270 |
| Mallory-Weiss syndrome | 10026712 |
| Mediastinal haematoma | 10049941 |
| Mediastinal haemorrhage | 10056343 |
| Medical device site bruise | 10075570 |
| Medical device site haematoma | 10075577 |
| Medical device site haemorrhage | 10075578 |
| Melaena | 10073378 |
| Melaena neonatal | 10027141 |
| Meningorrhagia | 10052593 |
| Menometrorrhagia | 10027295 |
| Menorrhagia | 10027313 |
| Mesenteric haematoma | 10071557 |
| Mesenteric haemorrhage | 10060717 |
| Metrorrhagia | 10027514 |
| Mouth haemorrhage | 10028024 |
| Mucocutaneous haemorrhage | 10076048 |
| Mucosal haemorrhage | 10061298 |
| Muscle contusion | 10070757 |
| Muscle haemorrhage | 10070757 |
| Myocardial haemorrhage | 10048849 |




| Myocardial rupture | 10028604 |
|---------------------------------------|----------|
| Naevus haemorrhage | 10062955 |
| Nail bed bleeding | 10048891 |
| Nasal septum haematoma | 10075027 |
| Neonatal gastrointestinal haemorrhage | 10074159 |
| Nephritis haemorrhagic | 10029132 |
| Nipple exudate bloody | 10029418 |
| Ocular retrobulbar haemorrhage | 10057571 |
| Oesophageal haemorrhage | 10030172 |
| Oesophageal intramural haematoma | 10077486 |
| Oesophageal ulcer haemorrhage | 10030202 |
| Oesophageal varices haemorrhage | 10030210 |
| Oesophagitis haemorrhagic | 10030219 |
| Optic disc haemorrhage | 10030919 |
| Optic nerve sheath haemorrhage | 10030941 |
| Oral blood blister | 10076590 |
| Oral contusion | 10078170 |
| Oral mucosa haematoma | 10074779 |
| Oral purpura | 10083533 |
| Orbital haematoma | 10083565 |
| Orbital haemorrhage | 10031045 |
| Osteorrhagia | 10051937 |
| Ovarian haematoma | 10033263 |
| Ovarian haemorrhage | 10065741 |
| Palpable purpura | 10056872 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic pseudocyst haemorrhage | 10083813 |
| Pancreatitis haemorrhagic | 10033650 |
| Papillary muscle haemorrhage | 10059164 |
| Paranasal sinus haematoma | 10069702 |
| Paranasal sinus haemorrhage | 10080108 |
| Parathyroid haemorrhage | 10059051 |
| Parotid gland haemorrhage | 10051166 |
| Pelvic haematoma | 10054974 |
| Pelvic haematoma obstetric | 10034248 |
| Pelvic haemorrhage | 10063678 |
| Penile contusion | 10073352 |
| Penile haematoma | 10070656 |
| Penile haemorrhage | 10034305 |
| Peptic ulcer haemorrhage | 10034344 |
| Pericardial haemorrhage | 10034476 |
| Perineal haematoma | 10034520 |
| Periorbital haematoma | 10034544 |
| Periorbital haemorrhage | 10071697 |
| Periosteal haematoma | 10077341 |
| Peripartum haemorrhage | 10072693 |
| Peripheral artery aneurysm rupture | 10079908 |




| Peripheral artery haematoma | 10081077 |
|----------------------------------------------------|----------|
| Peritoneal haematoma | 10058095 |
| Periventricular haemorrhage neonatal | 10076706 |
| Petechiae | 10034754 |
| Pharyngeal contusion | 10083176 |
| Pharyngeal haematoma | 10068121 |
| Pharyngeal haemorrhage | 10034827 |
| Pituitary apoplexy | 10056447 |
| Pituitary haemorrhage | 10049760 |
| Placenta praevia haemorrhage | 10035121 |
| Polymenorrhagia | 10064050 |
| Post abortion haemorrhage | 10036246 |
| Post procedural contusion | 10073353 |
| Post procedural haematoma | 10063188 |
| Post procedural haematuria | 10066225 |
| Post procedural haemorrhage | 10051077 |
| Post transfusion purpura | 10072265 |
| Postmenopausal haemorrhage | 10055870 |
| Postpartum haemorrhage | 10036417 |
| Post-traumatic punctate intraepidermal haemorrhage | 10071639 |
| Premature separation of placenta | 10036608 |
| Procedural haemorrhage | 10071229 |
| Proctitis haemorrhagic | 10036778 |
| Prostatic haemorrhage | 10036960 |
| Pulmonary alveolar haemorrhage | 10037313 |
| Pulmonary contusion | 10037370 |
| Pulmonary haematoma | 10054991 |
| Pulmonary haemorrhage | 10037394 |
| Pulmonary haemorrhage neonatal | 10082194 |
| Puncture site bruise | 10082035 |
| Puncture site haematoma | 10081957 |
| Puncture site haemorrhage | 10051101 |
| Purpura | 10037549 |
| Purpura fulminans | 10037556 |
| Purpura neonatal | 10037557 |
| Purpura non-thrombocytopenic | 10057739 |
| Purpura senile | 10037560 |
| Putamen haemorrhage | 10058940 |
| Radiation associated haemorrhage | 10072281 |
| Rectal haemorrhage | 10038063 |
| Rectal ulcer haemorrhage | 10038081 |
| Renal artery perforation | 10075737 |
| Renal cyst haemorrhage | 10059846 |
| Renal haematoma | 10038459 |
| Renal haemorrhage | 10038460 |
| Respiratory tract haemorrhage | 10038727 |
| Respiratory tract haemorrhage neonatal | 10038728 |




| | 10070101 |
|------------------------------------|-----------|
| Retinal aneurysm rupture | 10079121 |
| Retinal haemorrhage | 10038867 |
| Retinopathy haemorrhagic | 10051447 |
| Retroperitoneal haematoma | 10058360 |
| Retroperitoneal haemorrhage | 10038980 |
| Retroplacental haematoma | 10054798 |
| Ruptured cerebral aneurysm | 10039330 |
| Scleral haemorrhage | 10050508 |
| Scrotal haematocoele | 10061517 |
| Scrotal haematoma | 10039749 |
| | 10039749 |
| Scrotal haemorrhage | |
| Shock haemorrhagic | 10049771 |
| Skin haemorrhage | 10064265 |
| Skin neoplasm bleeding | 10060712 |
| Skin ulcer haemorrhage | 10050377 |
| Small intestinal haemorrhage | 10052535 |
| Small intestinal ulcer haemorrhage | 10061550 |
| Soft tissue haemorrhage | 10051297 |
| Spermatic cord haemorrhage | 10065742 |
| Spinal cord haematoma | 10076051 |
| Spinal cord haemorrhage | 10048992 |
| Spinal epidural haematoma | 10050162 |
| Spinal epidural haemorrhage | 10049236 |
| Spinal subarachnoid haemorrhage | 10073564 |
| Spinal subdural haematoma | 10050164 |
| Spinal subdural haemorrhage | 10073563 |
| Spleen contusion | 10073533 |
| Splenic artery perforation | 10075738 |
| Splenic haematoma | 10075756 |
| | 10041647 |
| Splenic haemorrhage | |
| Splenic varices haemorrhage | 10068662 |
| Splinter haemorrhages | 10041663 |
| Spontaneous haematoma | 10065304 |
| Spontaneous haemorrhage | 10074557 |
| Stoma site haemorrhage | 10074508 |
| Stomatitis haemorrhagic | 10042132 |
| Subarachnoid haematoma | 10076701 |
| Subarachnoid haemorrhage | 10042316 |
| Subarachnoid haemorrhage neonatal | 10042317 |
| Subcapsular hepatic haematoma | 10083383 |
| Subcapsular renal haematoma | 10083385 |
| Subcapsular splenic haematoma | 10083384 |
| Subchorionic haematoma | 10072596 |
| Subchorionic haemorrhage | 10071010 |
| Subclavian artery perforation | 10075740 |
| Subclavian vein perforation | 10075743 |
| Subcutaneous haematoma | 10073743 |
| DOCCHARCOUS HACHIAUDHA | TOUT LUTY |




| Subdural haematoma | 10042361 |
|---------------------------------------------------|----------|
| Subdural haematoma evacuation | 10042363 |
| Subdural haemorrhage | 10042364 |
| Subdural haemorrhage neonatal | 10042365 |
| Subendocardial haemorrhage | 10082459 |
| Subgaleal haematoma | 10069510 |
| Subgaleal haemorrhage | 10080900 |
| Subretinal haematoma | 10071935 |
| Superior vena cava perforation | 10075741 |
| Testicular haemorrhage | 10051877 |
| Thalamus haemorrhage | 10058939 |
| Third stage postpartum haemorrhage | 10043449 |
| Thoracic haemorrhage | 10062744 |
| Thrombocytopenic purpura | 10043561 |
| Thrombotic thrombocytopenic purpura | 10043648 |
| Thyroid haemorrhage | 10064224 |
| Tongue haematoma | 10043959 |
| Tongue haemorrhage | 10049870 |
| Tonsillar haemorrhage | 10057450 |
| Tooth pulp haemorrhage | 10072228 |
| Tooth socket haemorrhage | 10064946 |
| Tracheal haemorrhage | 10062543 |
| Traumatic haematoma | 10044522 |
| Traumatic haemorrhage | 10053476 |
| Traumatic haemothorax | 10074487 |
| Traumatic intracranial haematoma | 10079013 |
| Traumatic intracranial haemorrhage | 10079013 |
| Tumour haemorrhage | 10001387 |
| Ulcer haemorrhage | 10049730 |
| | 10061577 |
| Umbilical cord haemorrhage<br>Umbilical haematoma | |
| | 10068712 |
| Umbilical haemorrhage | 10045455 |
| Upper gastrointestinal haemorrhage | 10046274 |
| Ureteric haemorrhage | 10065743 |
| Urethral haemorrhage | 10049710 |
| Urinary bladder haematoma | 10083358 |
| Urinary bladder haemorrhage | 10046528 |
| Urogenital haemorrhage | 10050058 |
| Uterine haematoma | 10063875 |
| Uterine haemorrhage | 10046788 |
| Vaccination site bruising | 10069484 |
| Vaccination site haematoma | 10069472 |
| Vaccination site haemorrhage | 10069475 |
| Vaginal haematoma | 10046909 |
| Vaginal haemorrhage | 10046910 |
| Varicose vein ruptured | 10046999 |
| Vascular access site bruising | 10077767 |




| | Vascular access site haematoma | 10077647 |
|------------------|-----------------------------------------------|----------|
| | Vascular access site haemorrhage | 10077643 |
| | Vascular access site rupture | 10077652 |
| | Vascular anastomotic haemorrhage | 10084092 |
| | Vascular graft haemorrhage | 10077721 |
| | Vascular pseudoaneurysm ruptured | 10053949 |
| | Vascular purpura | 10047097 |
| | Vascular rupture | 10053649 |
| | Vein rupture | 10077110 |
| | Venous haemorrhage | 10065441 |
| | Venous perforation | 10075733 |
| | Ventricle rupture | 10047279 |
| | Vertebral artery perforation | 10075735 |
| | Vessel puncture site bruise | 10063881 |
| | Vessel puncture site haematoma | 10065902 |
| | Vessel puncture site haemorrhage | 10054092 |
| | Vitreous haematoma | 10071936 |
| | Vitreous haemorrhage | 10047655 |
| | Vulval haematoma | 10047756 |
| | Vulval haematoma evacuation | 10047757 |
| | Vulval haemorrhage | 10063816 |
| | Withdrawal bleed | 10047998 |
| | Wound haematoma | 10071504 |
| | Wound haemorrhage | 10051373 |
| Cholestasis and | Bilirubin excretion disorder | 10061009 |
| jaundice of | Cholaemia | 10048611 |
| hepatic origin | Cholestasis | 10008635 |
| | Cholestatic liver injury | 10067969 |
| | Cholestatic pruritus | 10064190 |
| | Drug-induced liver injury | 10072268 |
| | Hepatitis cholestatic | 10019754 |
| | Hyperbilirubinaemia | 10020578 |
| | Icterus index increased | 10021209 |
| | Jaundice | 10023126 |
| | Jaundice cholestatic | 10023129 |
| | Jaundice hepatocellular | 10023136 |
| | Mixed liver injury | 10066758 |
| | Ocular icterus | 10058117 |
| | Parenteral nutrition associated liver disease | 10074151 |
| Hepatic failure, | Acquired hepatocerebral degeneration | 10080860 |
| fibrosis and | Acute hepatic failure | 10000804 |
| cirrhosis and | Acute on chronic liver failure | 10077305 |
| other liver | Acute yellow liver atrophy | 10070815 |
| damage-related | Ascites | 10003445 |
| conditions | Asterixis | 10003547 |
| | Bacterascites | 10068547 |
| | Biliary cirrhosis | 10004659 |




| Biliary fibrosis | 10004664 |
|----------------------------------------------------|----------|
| | 10082480 |
| Cardiohepatic syndrome | |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10001937 |
| Hepatic calcification | 10015037 |
| Hepatic cirrhosis | 10003274 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Immune-mediated cholangitis | 10083406 |
| Immune-mediated hepatic disorder | 10083521 |
| Intestinal varices | 10083521 |
| Intestinal varices Intestinal varices haemorrhage | 10071302 |
| Liver dialysis | 10076640 |
| Liver disorder | 10070040 |
| Liver injury | 10067125 |
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |




| | Minimal hepatic encephalopathy | 10076204 |
|-----------------|--------------------------------------------|----------|
| | Mixed liver injury | 10070204 |
| | | 1 |
| | Nodular regenerative hyperplasia | 10051081 |
| | Nonalcoholic fatty liver disease | 10082249 |
| | Non-alcoholic steatohepatitis | 10053219 |
| | Non-cirrhotic portal hypertension | 10077259 |
| | Oedema due to hepatic disease | 10049631 |
| | Oesophageal varices haemorrhage | 10030210 |
| | Peripancreatic varices | 10073215 |
| | Portal fibrosis | 10074726 |
| | Portal hypertension | 10036200 |
| | Portal hypertensive colopathy | 10079446 |
| | Portal hypertensive enteropathy | 10068923 |
| | Portal hypertensive enteropathy | 10050897 |
| | Portal vein cavernous transformation | 10073979 |
| | Portal vein dilatation | 10073209 |
| | | 10073209 |
| | Portopulmonary hypertension | |
| | Primary biliary cholangitis | 10080429 |
| | Regenerative siderotic hepatic nodule | 10080679 |
| | Renal and liver transplant | 10052279 |
| | Retrograde portal vein flow | 10067338 |
| | Reye's syndrome | 10039012 |
| | Reynold's syndrome | 10070953 |
| | Splenic varices | 10067823 |
| | Splenic varices haemorrhage | 10068662 |
| | Steatohepatitis | 10076331 |
| | Subacute hepatic failure | 10056956 |
| | Sugiura procedure | 10083010 |
| | Varices oesophageal | 10056091 |
| | Varicose veins of abdominal wall | 10072284 |
| | White nipple sign | 10078438 |
| Hepatitis, non- | Acute graft versus host disease in liver | 10066263 |
| infectious | | |
| intectious | Allergic hepatitis | 10071198 |
| | Alloimmune hepatitis | 10080576 |
| | Autoimmune hepatitis | 10003827 |
| | Chronic graft versus host disease in liver | 10072160 |
| | Chronic hepatitis | 10008909 |
| | Graft versus host disease in liver | 10064676 |
| | Hepatitis | 10019717 |
| | Hepatitis acute | 10019727 |
| | Hepatitis cholestatic | 10019754 |
| | Hepatitis chronic active | 10019755 |
| | Hepatitis chronic persistent | 10019759 |
| | Hepatitis fulminant | 10019772 |
| | Hepatitis toxic | 10019795 |
| | Immune-mediated hepatitis | 10078962 |
| | Ischaemic hepatitis | 10073902 |
| | Ischaeme nepautis | 10023023 |




| | Lupus hepatitis | 10067737 |
|---|---|---|
| | Non-alcoholic steatohepatitis | 10057737 |
| | | 10053219 |
| | Radiation hepatitis | |
| T : 1-4-1 | Steatohepatitis | 10076331 |
| Liver related | Alanine aminotransferase abnormal | 10001547 |
| investigations, | Alanine aminotransferase increased | 10001551 |
| signs and | Ammonia abnormal | 10001942 |
| symptoms | Ammonia increased | 10001946 |
| | Ascites | 10003445 |
| | Aspartate aminotransferase abnormal | 10003477 |
| | Aspartate aminotransferase increased | 10003481 |
| | AST/ALT ratio abnormal | 10082832 |
| | Bacterascites | 10068547 |
| | Bile output abnormal | 10051344 |
| | Bile output decreased | 10051343 |
| | Biliary ascites | 10074150 |
| | Bilirubin conjugated abnormal | 10067718 |
| | Bilirubin conjugated increased | 10004685 |
| | Bilirubin urine present | 10077356 |
| | Biopsy liver abnormal | 10004792 |
| | Blood bilirubin abnormal | 10058477 |
| | Blood bilirubin increased | 10005364 |
| | Blood bilirubin unconjugated increased | 10005370 |
| | Bromosulphthalein test abnormal | 10006408 |
| | Child-Pugh-Turcotte score abnormal | 10077020 |
| | Child-Pugh-Turcotte score increased | 10068287 |
| | Computerised tomogram liver abnormal | 10078360 |
| | Congestive hepatopathy | 10084058 |
| | Foetor hepaticus | 10052554 |
| | Galactose elimination capacity test abnormal | 10052554 |
| | Galactose elimination capacity test abnormal | 10059710 |
| | Gamma-glutamyltransferase abnormal | 10039712 |
| | Gamma-glutamyltransferase increased | 10017688 |
| | Guanase increased | |
| | | 10051333<br>10019621 |
| | Hepaplastin abnormal | |
| | Hepaplastin decreased | 10019622 |
| | Hepatic artery flow decreased | 10068997 |
| | Hepatic enzyme abnormal | 10062685 |
| | Hepatic enzyme decreased | 10060794 |
| | Hepatic enzyme increased | 10060795 |
| | Hepatic function abnormal | 10019670 |
| | Hepatic hydrothorax | 10067365 |
| | Hepatic hypertrophy | 10076254 |
| | Hepatic mass | 10057110 |
| | Hepatic pain | 10019705 |
| | Hepatic sequestration | 10066244 |
| | Hepatic vascular resistance increased | 10068358 |




| | Hepatic venous pressure gradient abnormal | 10083172 |
|---|---|---|
| | Hepatic venous pressure gradient increased | 10083172 |
| | Hepatobiliary scan abnormal | 1 |
| | | 10066195 |
| | Hepatomegaly | 10019842 |
| | Hepatosplenomegaly | 10019847 |
| | Hyperammonaemia | 10020575 |
| | Hyperbilirubinaemia | 10020578 |
| | Hypercholia | 10051924 |
| | Hypertransaminasaemia | 10068237 |
| | Kayser-Fleischer ring | 10023321 |
| | Liver function test abnormal | 10024690 |
| | Liver function test decreased | 10077677 |
| | Liver function test increased | 10077692 |
| | Liver induration | 10052550 |
| | Liver palpable | 10075895 |
| | Liver scan abnormal | 10061947 |
| | Liver tendemess | 10024712 |
| | Magnetic resonance imaging liver abnormal | 10083123 |
| | Magnetic resonance proton density fat fraction measurement | 10082443 |
| | Mitochondrial aspartate aminotransferase increased | 10064712 |
| | Molar ratio of total branched-chain amino acid to tyrosine | 10066869 |
| | Oedema due to hepatic disease | 10049631 |
| | Perihepatic discomfort | 10054125 |
| | Retrograde portal vein flow | 10067338 |
| | Total bile acids increased | 10064558 |
| | Transaminases abnormal | 10062688 |
| | Transaminases increased | 10054889 |
| | Ultrasound liver abnormal | 10045428 |
| | Urine bilirubin increased | 10050792 |
| | White nipple sign | 10078438 |
| | X-ray hepatobiliary abnormal | 10056536 |
| Hypertension | Accelerated hypertension | 10000358 |
| | Blood pressure ambulatory increased | 10005732 |
| | Blood pressure diastolic increased | 10005739 |
| | Blood pressure inadequately controlled | 10051128 |
| | Blood pressure increased | 10005750 |
| | Blood pressure management | 10063926 |
| | Blood pressure orthostatic increased | 10053355 |
| | Blood pressure systolic increased | 10005760 |
| | Catecholamine crisis | 10081751 |
| | Dialysis induced hypertension | 10063067 |
| | Diastolic hypertension | 10012758 |
| | Eclampsia | 10014129 |
| | Endocrine hypertension | 10057615 |
| | Essential hypertension | 10015488 |
| | Gestational hypertension | 10070538 |
| | HELLP syndrome | 10049058 |
| | I DO STATE OF THE | 10012030 |




| | Hyperaldosteronism | 10020571 |
|-------------|----------------------------------------|----------|
| | Hypertension | 10020772 |
| | Hypertension neonatal | 10049781 |
| | Hypertensive angiopathy | 10049781 |
| | Hypertensive cardiomegaly | 10039238 |
| | | 1 |
| | Hypertensive cardiomyopathy | 10058222 |
| | Hypertensive cerebrovascular disease | 10077000 |
| | Hypertensive crisis | 10020802 |
| | Hypertensive emergency | 10058179 |
| | Hypertensive encephalopathy | 10020803 |
| | Hypertensive end-organ damage | 10079496 |
| | Hypertensive heart disease | 10020823 |
| | Hypertensive nephropathy | 10055171 |
| | Hypertensive urgency | 10058181 |
| | Labile hypertension | 10049079 |
| | Malignant hypertension | 10025600 |
| | Malignant hypertensive heart disease | 10025603 |
| | Malignant renal hypertension | 10026674 |
| | Maternal hypertension affecting foetus | 10026924 |
| | Mean arterial pressure increased | 10026985 |
| | Metabolic syndrome | 10052066 |
| | Neurogenic hypertension | 10067598 |
| | Orthostatic hypertension | 10065508 |
| | Page kidney | 10076704 |
| | Postoperative hypertension | 10050631 |
| | Pre-eclampsia | 10036485 |
| | Prehypertension | 10050485 |
| | Procedural hypertension | 10062886 |
| | Renal hypertension | 10038464 |
| | Renal sympathetic nerve ablation | 10074864 |
| | Renovascular hypertension | 10038562 |
| | Retinopathy hypertensive | 10038926 |
| | Secondary aldosteronism | 10039808 |
| | Secondary hypertension | 10039834 |
| | Supine hypertension | 10078932 |
| | Systolic hypertension | 10042957 |
| | Withdrawal hypertension | 10048007 |
| Proteinuria | Albumin globulin ratio increased | 10001567 |
| | Albumin urine present | 10001582 |
| | Albuminuria | 10001580 |
| | Bence Jones protein urine present | 10053112 |
| | Bence Jones proteinuria | 10004231 |
| | Beta 2 microglobulin urine increased | 10004501 |
| | Globulinuria | 10018352 |
| | Microalbuminuria | 10027525 |
| | Myoglobinuria | 10028629 |
| | Orthostatic proteinuria | 10031129 |
| | отпознае реченина | 10031123 |




| | Protein urine | 10037018 |
|-------------|-----------------------------------------------------|----------|
| | Protein urine present | 10053123 |
| | Proteinuria | 10037032 |
| | Urine albumin/creatinine ratio increased | 10053541 |
| | Urine protein/creatinine ratio abnormal | 10053539 |
| | Urine protein/creatinine ratio increased | 10053538 |
| Thyroid | Basedow's disease | 10004161 |
| dysfunction | Endocrine ophthalmopathy | 10060742 |
| | Exophthalmos | 10015683 |
| | Hashitoxicosis | 10067873 |
| | Hyperthyroidism | 10020850 |
| | Immune-mediated hyperthyroidism | 10083517 |
| | Inappropriate thyroid stimulating hormone secretion | 10075007 |
| | Malignant exophthalmos | 10075386 |
| | Marine Lenhart syndrome | 10068828 |
| | Primary hyperthyroidism | 10075899 |
| | Secondary hyperthyroidism | 10053260 |
| | Thyroid dermatopathy | 10069771 |
| | Thyroid tuberculosis | 10043774 |
| | Thyrotoxic cardiomyopathy | 10075043 |
| | Thyrotoxic crisis | 10043786 |
| | Thyrotoxic myopathy | 10043780 |
| | Thyrotoxic periodic paralysis | 10081324 |
| | | 100.5700 |
| | Toxic goitre | 10075050 |
| | Toxic nodular goitre | 10044242 |
| | Anti-thyroid antibody | 10060325 |
| | Anti-thyroid antibody positive | 10060310 |
| | Antithyroid arthritis syndrome | 10073029 |
| | Autoimmune thyroid disorder | 10079165 |
| | Autoimmune thyroiditis | 10049046 |
| | Biopsy thyroid gland abnormal | 10004889 |
| | Blood thyroid stimulating hormone abnormal | 10005830 |
| | Blood thyroid stimulating hormone decreased | 10005832 |
| | Blood thyroid stimulating hormone increased | 10005833 |
| | Butanol-extractable iodine decreased | 10006818 |
| | Butanol-extractable iodine increased | 10006819 |
| | Congenital thyroid disorder | 10076602 |
| | Euthyroid sick syndrome | 10015549 |
| | Free thyroxine index abnormal | 10050747 |
| | Free thyroxine index decreased | 10050748 |
| | Free thyroxine index increased | 10050749 |
| | Gamma radiation therapy to thyroid | 10017685 |
| | Goitre | 10018498 |
| | Hashimoto's encephalopathy | 10069432 |
| | Immune-mediated thyroiditis | 10083071 |
| | Infectious thyroiditis | 10071250 |
| | Iodine uptake abnormal | 10022918 |
| | Produc abrance activities | 10022310 |




| T-di | 1000000 |
|---------------------------------------------------|----------|
| Iodine uptake decreased | 10022920 |
| Iodine uptake increased | 10022922 |
| Orbital decompression | 10072141 |
| Photon radiation therapy to thyroid | 10034957 |
| Polyglandular autoimmune syndrome type II | 10036073 |
| Polyglandular autoimmune syndrome type III | 10064115 |
| Protein bound iodine decreased | 10037001 |
| Protein bound iodine increased | 10037002 |
| Radioactive iodine therapy | 10037784 |
| Radiotherapy to thyroid | 10062098 |
| Reverse tri-iodothyronine decreased | 10060307 |
| Reverse tri-iodothyronine increased | 10060306 |
| Silent thyroiditis | 10079012 |
| Thyreostatic therapy | 10065359 |
| Thyroglobulin absent | 10054025 |
| Thyroglobulin decreased | 10054011 |
| Thyroglobulin increased | 10054010 |
| Thyroglobulin present | 10054024 |
| Thyroid disorder | 10043709 |
| Thyroid dysfunction in pregnancy | 10056525 |
| Thyroid electron radiation therapy | 10043722 |
| Thyroid function test abnormal | 10043730 |
| Thyroid gland scan abnormal | 10062149 |
| Thyroid hemiagenesis | 10077609 |
| Thyroid hormone replacement therapy | 10068076 |
| Thyroid hormones increased | 10063161 |
| Thyroid operation | 10062126 |
| Thyroid pain | 10043757 |
| Thyroid releasing hormone challenge test abnormal | 10043764 |
| Thyroid stimulating immunoglobulin increased | 10071389 |
| Thyroid therapy | 10065358 |
| Thyroidectomy | 10062127 |
| Thyroiditis | 10043778 |
| Thyroiditis acute | 10043780 |
| Thyroiditis chronic | 10043781 |
| Thyroiditis fibrous chronic | 10043782 |
| Thyroiditis subacute | 10043784 |
| Thyroxin binding globulin abnormal | 10051423 |
| Thyroxin binding globulin decreased | 10051421 |
| Thyroxin binding globulin increased | 10051420 |
| Thyroxine abnormal | 10043814 |
| Thyroxine decreased | 10043816 |
| Thyroxine free abnormal | 10055158 |
| Thyroxine free decreased | 10055162 |
| Thyroxine free increased | 10055163 |
| Thyroxine increased | 10043818 |
| Thyroxine therapy | 10052702 |
| AMIANUM MARKET | 10052702 |




| Tri-iodothyronine abnormal | 10044592 |
|--------------------------------------------|----------|
| | 10044594 |
| Tri-iodothyronine decreased | 2001.221 |
| Tri-iodothyronine free abnormal | 10053794 |
| Tri-iodothyronine free decreased | 10053791 |
| Tri-iodothyronine free increased | 10053790 |
| Tri-iodothyronine free normal | 10053793 |
| Tri-iodothyronine increased | 10044596 |
| Tri-iodothyronine uptake abnormal | 10062215 |
| Tri-iodothyronine uptake decreased | 10044601 |
| Tri-iodothyronine uptake increased | 10044602 |
| Ultrasound thyroid abnormal | 10060987 |
| X-ray therapy to thyroid | 10048207 |
| Autoimmune hypothyroidism | 10076644 |
| Congenital hypothyroidism | 10010510 |
| Generalised resistance to thyroid hormone | 10018096 |
| Hypothyroidic goitre | 10059844 |
| Hypothyroidism | 10021114 |
| Immune-mediated hypothyroidism | 10083075 |
| Myxoedema | 10028665 |
| Myxoedema coma | 10060819 |
| Post procedural hypothyroidism | 10065306 |
| Primary hypothyroidism | 10036697 |
| Secondary hypothyroidism | 10039840 |
| Tertiary hypothyroidism | 10043289 |
| Thyroid atrophy | 10043693 |
| Thyroid stimulating hormone deficiency | 10078564 |
| Transient hypothyroxinaemia of prematurity | 10075901 |
| Atrophic thyroiditis | 10077172 |

# **Certificate Of Completion**

Envelope Id: PPD

Subject: Complete with DocuSign: Hutchison 2015-012-00US1 SAP Final V2.2\_20221104.docx

Project Code (Enter 0 for non-billable projects): PPD

IQVIA ID (Login ID): PPD

Business Unit:

DSSR

Source Envelope: Document Pages: 70

Certificate Pages: 5 AutoNav: Enabled

Envelopeld Stamping: Disabled Time Zone: (UTC+08:00) Taipei

Signatures: 3 Initials: 0

Envelope Originator:

Status: Completed

PPD

One IMS Way

Plymouth Meeting, 19462

PPD

### Record Tracking

Status: Original

06-Nov-2022 | 18:28

Holder: PPD

Location: DocuSign

### Signer Events

### PPD

Security Level: Email, Account Authentication (Required)

Signature

PPD

**Timestamp** 

Sent: 06-Nov-2022 | 18:40 Viewed: 07-Nov-2022 | 09:54 Signed: 07-Nov-2022 | 10:59

Signature Adoption: Pre-selected Style

Signature ID:

PPD

Using IP Address: PPD

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

# Electronic Record and Signature Disclosure:

Accepted: 07-Nov-2022 | 09:54 ID: PPD

PPD

Security Level: Email, Account Authentication (Required)

PPD

Sent: 07-Nov-2022 | 10:59 Viewed: 07-Nov-2022 | 17:34 Signed: 07-Nov-2022 | 17:35

Signature Adoption: Pre-selected Style

Signature ID:

PPD

Using IP Address: PPD

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

Electronic Record and Signature Disclosure:

Accepted: 28-Apr-2021 | 02:03

ID: PPD

Signer Events Signature Timestamp PPD Sent: 07-Nov-2022 | 17:35 PPD Viewed: 07-Nov-2022 | 19:26 Security Level: Email, Account Authentication Signed: 07-Nov-2022 | 19:27 (Required) Signature Adoption: Pre-selected Style Signature ID: PPD Using IP Address: PPD

> With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

Electronic Record and Signature Disclosure: Accepted: 07-Nov-2022 | 19:25 ID: PPD

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 06-Nov-2022 18:40<br>07-Nov-2022 19:26<br>07-Nov-2022 19:27<br>07-Nov-2022 19:27 |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

# Documents will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

# Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

# Consequences of Withdrawing Consent

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

### How to contact IQVIA:

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact

1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to compare to the compare of the compare

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

# 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to CCI

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

# 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to consent; or and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

# Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security<br>Settings: | Allow per session cookies |
| Mobile Signing: | Apple iOS 7.0 or above Android 4.0 or above |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.